

March 22, 2022

Clinicaltrials.gov

#### To Whom it May Concern:

Following please find the Statistical Analysis Plan (SAP) for the study titled "Randomized, Double-Blind, Sham-Controlled, Prospective, Multi-Center Pilot Study to Evaluate the Safety and Effectiveness of Duodenal Mucosal Resurfacing Using the Revita™ System in the Treatment of Type 2 Diabetes", version date 19May2020, NCT03653091.

Sincerely,

Docusigned by:

Sarah Hackett

FF259F44539D417...

Sarah Hackett Sr. Director of Clinical Operations Fractyl Health

# Statistical Analysis Plan



| Sponsor | Fractyl Laboratories, Inc. |
|---|---|
| Protocol Title: | Randomized, Double-Blind, Sham-Controlled, Prospective, Multi-Center Pilot Study to Evaluate the Safety and Effectiveness of Duodenal Mucosal Resurfacing Using the Revita <sup>TM</sup> System in the Treatment of Type 2 Diabetes |
| Protocol Number: | C-40000 |
| Premier Research PCN: | FRAC8070 |
| Document Version: | Version 1.0 |
| Document Date: | 19-May-2020 |

## Approvals

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| Lead<br>Biostatistician | Print Name: Adrienne Kuxhausen, M.S. Sign Name: DocuSigned by: Marienne kuxhausen Signer Name: Adrienne Kuxhausen Signing Reason: I am the author of this document Signing Time: 19-May-2020 18:06:45 EDT 6E6B87C6B98740819F26B8D5A7D662CF | |
| Premier Statistical<br>Reviewer | Print Name: Valerie H. Smith, MStat Sign Name: DocuSigned by: Valerie Smith Signer Name: Valerie Smith Signing Reason: I have reviewed this document Signing Time: 19-May-2020 18:42:14 EDT 882C53F2B5164EEAA9FA446FC310D506 | |



| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| Fractyl<br>Representative<br>(Senior<br>Biostatistician) | Print Name: Vijeta Bhambhani, M.S, MPH. Sign Name: DocuSigned by: Vijeta Bhambhani Signer Name: Vijeta Bhambhani Signing Reason: I approve this document Signing Time: 19-May-2020 15:44:47 PDT 57D62E5BA6394781AA7C96A3CE5C9599 | |
| Fractyl<br>Representative<br>(Chief Medical<br>Officer) | Print Name: Juan Carlos Lopez-Talavera, MD, PhD Sign Name: DocuSigned by: Juan Carlos Lopez-Talavera Signer Name: Juan Carlos Lopez-Talavera Signing Reason: I have reviewed this document Signing Time: 19-May-2020 18:42:44 EDT 03D500585DE143C2880D2B2392934776 | |





## **Document History**

Not applicable.



## **Table of Contents**

| Ov | erview | 7 |
|---|---|---|
| Stu | ndy Objectives and Endpoints | 7 |
| 2.1. | Study Objectives | 7 |
| 2.2. | Study Endpoints | 7 |
| 2.2.1. | Safety Endpoints | 7 |
| 2.2.2. | Efficacy Endpoints | 8 |
| 2.2.2.3 | Additional Efficacy Endpoint | 8 |
| Ov | rerall Study Design and Plan | 8 |
| 3.1. | Overall Design | 9 |
| 3.2. | Sample Size and Power. | 9 |
| 3.3. | Study Population | 9 |
| 3.4. | Treatments Administered | 9 |
| 3.5. | Method of Assigning Subjects to Treatment Groups | 10 |
| 3.6. | Blinding and Unblinding. | 10 |
| 3.7. | Schedule of Events | 11 |
| Sta | tistical Analysis and Reporting | 19 |
| 4.1. | Introduction | 19 |
| 4.2. | Interim Analysis and Data Monitoring | 19 |
| 4.2.1. | Clinical Events Committee | 20 |
| 4.2.2. | Data Monitoring Committee | 20 |
| An | alysis Populations | 21 |
| Ge | neral Issues for Statistical Analysis | 22 |
| 6.1. | Statistical Definitions and Algorithms | 22 |
| 6.1.1. | Baseline | 22 |
| 6.1.2. | Adjustments for Covariates. | 22 |
| 6.1.3. | Multiple Comparisons | 22 |
| 6.1.4. | Handling of Dropouts or Missing Data | 22 |
| 6.1.5. | Analysis Visit Windows | 22 |
| 6.1.6. | Pooling of Sites | 23 |
| 6.1.7. | Derived Variables | 23 |
| 6.1.8. | Data Adjustments/Handling/Conventions | 26 |
| Stu | ndy Subjects and Demographics | 27 |
| 7.1. | Disposition of Subjects and Withdrawals | 27 |
| 7.2. | Protocol Violations and Deviations | 27 |
| 7.3. | Demographics and Other Baseline Characteristics | 28 |
| | Stu 2.1. 2.2. 2.2.1. 2.2.2. 3.3. Ov 3.1. 3.2. 3.3. 3.4. 3.5. 3.6. 3.7. Sta 4.1. 4.2. 4.2.1. 4.2.2. An Ge 6.1. 6.1.1. 6.1.2. 6.1.3. 6.1.4. 6.1.5. 6.1.6. 6.1.7. 6.1.8. Stu 7.1. 7.2. | Study Objectives and Endpoints 2.1. Study Objectives 2.2. Study Endpoints 2.2.1. Safety Endpoints 2.2.2. Efficacy Endpoints 2.2.2. Efficacy Endpoints 2.2.2.3. Additional Efficacy Endpoint Overall Study Design and Plan 3.1. Overall Design 3.2. Sample Size and Power 3.3. Study Population 3.4. Treatments Administered 3.5. Method of Assigning Subjects to Treatment Groups 3.6. Blinding and Unblinding 3.7. Schedule of Events Statistical Analysis and Reporting 4.1. Introduction 4.2. Interim Analysis and Data Monitoring 4.2.1. Clinical Events Committee 4.2.2. Data Monitoring Committee 4.2.2. Data Monitoring Committee Analysis Populations General Issues for Statistical Analysis 6.1. Statistical Definitions and Algorithms 6.1.1. Baseline 6.1.2. Adjustments for Covariates 6.1.3. Multiple Comparisons 6.1.4. Handling of Dropouts or Missing Data 6.1.5. Analysis Visit Windows 6.1.6. Pooling of Sites 6.1.7. Derived Variables 6.1.8. Data Adjustments/Handling/Conventions Study Subjects and Demographics 7.1. Disposition of Subjects and Withdrawals 7.2. Protocol Violations and Deviations |





| | 7.4. | Exposure and Compliance | 28 |
|---|---|---|---|
| | 7.4.1. | Endoscopy and Endoscopic Evaluation | 28 |
| 8. | Ef | ficacy Analysis | 29 |
| | 8.1. | Primary Efficacy Analysis | 29 |
| | 8.2. | Secondary Efficacy Analysis | 29 |
| | 8.2.1. | HbA1c Over Time. | 29 |
| | 8.2.2. | Fasting Plasma Glucose (FPG) | 29 |
| | | Urine Albumin Creatinine Ratio (UACR) | |
| | 8.2.4. | Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) | 30 |
| | 8.3. | Additional Endpoints of Interest | 30 |
| | 8.3.1. | Short Form (36) Health Survey (SF-36) | 30 |
| | 8.3.2. | Patient Reported Outcomes Measurement Information System (PROMIS®) | 30 |
| 9. | Sa | fety and Tolerability Analysis | 30 |
| | 9.1. | Adverse Events | 31 |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 31 |
| | 9.1.2. | Deaths and Serious Adverse Events | 32 |
| | 9.1.3. | Other Significant Adverse Events | 32 |
| | 9.1.3. | . Unanticipated Adverse Device Effects (UADEs) | 32 |
| | 9.1.3.2 | 2. Adverse Events of Special Interest (AESIs) | 32 |
| | 9.2. | Clinical Laboratory Evaluations | 33 |
| | 9.3. | Vital Signs | 33 |
| | 9.4. | Electrocardiograms | 33 |
| | 9.5. | Further Safety Evaluations | 34 |
| | 9.5.1. | MRI Enterography | 34 |
| | 9.5.2. | Lifestyle Counseling and Evaluation | 34 |
| | 9.6. | Concomitant Medication | 34 |
| | 9.7. | Physical Exam. | 34 |
| 10. | Cł | anges from Planned Analysis | 34 |
| 11. | Ot | her Planned Analysis | 35 |
| 12. | Re | ferences | 36 |
| 13. | Ta | bles, Listings, and Figures | 36 |
| | 13.1. | Planned Table Descriptions | 37 |
| | 13.2. | Efficacy Data | 38 |
| | 13.3. | Safety Data | |
| | 13.4. | Planned Listing Descriptions | |
| 14. | Ta | bles, Listings, and Listing Shells | 46 |
| | 14.1. | Standard Layout for all Tables, Listings, and Figures | 46 |





| 48 |
|-----|
| 97 |
| 140 |
| 12 |
| 14 |
| 23 |
| 25 |
| 38 |
| 38 |
| 39 |
| 42 |
| 47 |
| 49 |



#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for Fractyl Laboratories Inc.'s protocol number C-40000 (Randomized, Double-Blind, Sham-Controlled, Prospective, Multi-Center Pilot Study to Evaluate the Safety and Effectiveness of Duodenal Mucosal Resurfacing Using the Revita<sup>TM</sup> System in the Treatment of Type 2 Diabetes), dated 29-Jan-2019 Version 2.0. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be documented in a supplemental SAP (drafted after lock) and clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to Fractyl's study C-40000.

#### 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

The study objectives are:

- To assess the safety of the Fractyl Revita<sup>TM</sup> System for the treatment of subjects with type 2 diabetes (T2D) suboptimally controlled on 2 to 3 oral antidiabetic medications (OADs)
- To assess the effect of Duodenal Mucosal Resurfacing (DMR) versus Sham procedures on glycemic endpoints 24 weeks after the procedure
- To assess the effect of DMR on glycemic endpoints 48 weeks after the procedure for durability of effect determination

#### 2.2. Study Endpoints

#### 2.2.1. Safety Endpoints

The safety endpoints of this study include the following:

• Event number and incidence of reported adverse events (AEs) and serious adverse events (SAEs), as well as device- and procedure-relatedness of AEs and SAEs, unanticipated adverse device effects (UADEs), and withdrawals due to AEs



Other safety endpoints include:

- Assessments including vital signs and weight, physical examinations, laboratory values, and electrocardiograms (ECGs)
- Duodenal biopsy samples for histological evidence of mucosal regrowth, inflammation and fibrosis
- Magnetic resonance imaging enterography (MRE) to assess thermal injury to the duodenum

#### 2.2.2. Efficacy Endpoints

#### 2.2.2.1. Primary Efficacy Endpoint

The primary efficacy endpoint of this study is HbA1c change from baseline to Week 24, DMR vs Sham.

#### 2.2.2.2. Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study include the following:

- (i) HbA1c change from baseline to Week 24 by visit over time, DMR vs. Sham
- (ii) Fasting plasma glucose (FPG) change from baseline to Week 24, DMR vs. Sham
- (iii) FPG change from baseline to Week 24 by visit over time, DMR vs. Sham
- (iv) Proportion of DMR-treated subjects with an HbA1c improvement from baseline at 24 weeks that maintain an HbA1c improvement at 48 weeks
- (v) Urine albumin-to-creatinine Ratio (UACR) change from baseline to Week 24, DMR vs. Sham
- (vi) Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) change from baseline to Week 24, DMR vs. Sham

#### 2.2.2.3. Additional Efficacy Endpoint

Additional efficacy endpoints of this study include the following:

- (i) HbA1c change from baseline to Week 48 by visit over time, DMR only
- (ii) FPG change from baseline to Week 48 by visit over time, DMR only
- (iii) UACR change from baseline to Week 48 by visit over time, DMR only
- (iv) ALT and AST change from baseline to Week 48 by visit over time, DMR only
- (v) HbA1c change from Week 24 (pre-DMR) in Sham cross-over group to Week 48
- (vi) FPG change from Week 24 (pre-DMR) in Sham cross-over group to Week 48
- (vii) Short Form (36) Health Survey Version 2 (SF-36) change from baseline at Week 24 (pre-assessments and endoscopy) vs Sham
- (viii) PROMIS® (Patient-Reported Outcomes Measurement Information System) change from baseline at Week 24 (pre-assessments and endoscopy) vs Sham

#### 3. Overall Study Design and Plan

The United States (US) pilot study is a prospective, randomized, double-blind (subject and endocrinologist), 24-week, Sham-controlled, multi-center, pilot trial in a maximum of 18 subjects with T2D suboptimally controlled on 2 to 3 OADs, one of which must be metformin.



Randomization will be 2:1 DMR treatment to Sham procedure. Total post-randomization study duration will be 48 weeks.

All eligible subjects will participate in a 4-week antidiabetic medication Run-In Period before randomization to the index procedure to assess stability of blood glucose control in conjunction with medication compliance and lifestyle (diet, exercise) counseling. OADs will be held constant from the start of the Run-In Period through Week 24, with protocol pre-specified treatment algorithms for hypoglycemia and hyperglycemia.

Following the medication Run-In Period, subjects will be scheduled for an endoscopic evaluation consisting of an assessment of the esophagus, stomach, duodenum and associated structures to ensure there are no conditions that would exclude the subject from having the index procedure (DMR or Sham).

Following confirmation of subject eligibility during the endoscopic evaluation, subjects will be randomized to receive the DMR or Sham procedure. Post-procedure, the subjects will be required to return for follow-up visits as per the visit schedule.

Both treatment groups will be followed up for a total of 48 weeks from the index procedure and will continue to receive lifestyle counseling through the end of the study. At the Week 24 visit, subjects will be unblinded and subjects randomized to the DMR treatment group will have an ablation site biopsy and will be followed for an additional 24 weeks. At the Week 24 visit, the Sham treatment group will be provided the opportunity to cross over to receive the DMR treatment. Sham subjects will then repeat all study visits from the DMR procedure through 24 weeks post crossover. Sham subjects that choose not to crossover and have the DMR treatment will be withdrawn from the study.

Subject follow up visits conducted by telephone will occur at 7 and 14 days and at Weeks 8, 15, 21, 30 and 42 post procedure. Subject follow up visits conducted in clinic will occur at Weeks 4, 12, 18, 24, 36 and 48 post procedure.

#### 3.1. Overall Design

#### 3.2. Sample Size and Power

The total study enrollment is planned to reach up to 18 subjects (12 DMR, 6 Sham). Sample size determination is based on the nature of this pilot study and not statistical considerations, therefore, this study is not statistically powered to demonstrate a statistically significant difference in effectiveness parameters between the treatment groups.

#### 3.3. Study Population

The protocol is written such that a maximum of 18 subjects at up to 6 study sites in the US will be enrolled into this clinical study. The clinical study population will be comprised of males and females, 28 - 65 years of age.

#### 3.4. Treatments Administered

The Fractyl Revita<sup>TM</sup> System consists of two main components: the Revita<sup>TM</sup> Catheter and a Console.

The Revita<sup>TM</sup> Catheter is a sterile, single use device that is delivered transorally over a guidewire into the duodenum using standard techniques, by a therapeutic endoscopist, and performs two



functions: 1) injects saline into the submucosa of the duodenum to create a thermal barrier while also lifting the mucosa with saline to create a more uniform surface for ablation; and 2) ablates the mucosal surface using heated water recirculating inside a balloon. The Revita<sup>TM</sup> catheter is placed in the proximal duodenum distal to the papilla.

The console is a reusable electro-mechanical piece of equipment and provides precisely controlled functionality to the catheter to perform the submucosal lift and hot fluid ablation steps of the procedure. The console is controlled by the user through the use of a software user interface monitor. Prior to use, the console is fitted with a sterile single use line set that serves as the pathway for the saline to be placed into the duodenal submucosa during the procedure.

The DMR procedure (mucosal lift and mucosal ablation) using the Revita<sup>TM</sup> System utilizes an over the wire endoscopic approach to ablate the duodenum. Using the console interface, the balloon is inflated and vacuum delivered to draw the intestinal mucosal tissue into the ports located on the balloon. The actuator on the handle is moved to advance the needle into the submucosal space within each of the ports. The console delivers saline colored with methylene blue or similar dye into the submucosa through the needles within the lumens of the catheter resulting in complete circumferential lift of the mucosa. Once complete, the ablation cycle is started and hot water is circulated into the balloon to complete an ablation of the previously expanded tissue. The balloon is deflated and the catheter repositioned distally to the next segment to be treated. The process of expansion, ablation and repositioning is repeated until the needed length is treated. A full DMR procedure is defined as 5 complete ablations representing 10 axial centimeters of circumferentially ablated tissue in the duodenum. The Revita<sup>TM</sup> catheter and endoscope are then removed.

The Sham procedure will consist of placing the Revita<sup>TM</sup> Catheter as described above into the duodenum for a minimum of 30 minutes and then removing it from the patient.

#### 3.5. Method of Assigning Subjects to Treatment Groups

Following confirmation of subject eligibility during the endoscopic evaluation, the subject will be randomized using electronic assignment via a web-based system at a 2:1 ratio to DMR procedure or Sham procedure.

#### 3.6. Blinding and Unblinding

In this study, the endocrinologist and the associated site personnel and the subjects will be blinded to the treatment through the Week 24 follow-up visit, as will the Sponsor study team (except the proctors and technicians who will be present at the procedure). While the endoscopist will not be blinded to individual treatments, he or she will be blinded to cohort level data and will not be responsible for the diabetes management of the subjects. At the Week 24 Visit, the subjects, the endocrinologist and the blinded study site staff, as well as the blinded Sponsor study team will be unblinded.

Subjects who received the Sham treatment will be offered the option to crossover and undergo the DMR procedure at the Week 24 Visit post randomization.

No study staff, associated hospital personnel, or study subjects will be informed of the randomization assignments until the scheduled time of unblinding at Week 24, and care will be taken to minimize the risk of inadvertent premature unblinding. The unblinding occurs after all assessments have been conducted at the Week 24 Visit.





#### 3.7. Schedule of Events

A detailed schedule of events for the DMR cases is provided in





## Table 1. A detailed schedule of events for the Sham cases is provided in



**premier** research

Table 1Table 2.



#### **Table 1: Schedule of Events—DMR Cases**

| Vis | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History &<br>Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pybri Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | DMR Procedure | Biopsy | Blinding Assessment | Lifestyle Counseling | SF-36 Questionnaire | PROMIS® Patient Reported<br>Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Diary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Screeni<br>ng<br>(Pre<br>Run-In) | | Х | X <sup>&amp;</sup> | | | х | х | х | | | | | | | | х | | | * | х | х |
| 2 | Baselin<br>e<br>(Post<br>Run-In) | Visit to<br>occur<br>4-6<br>weeks<br>after<br>Screeni<br>ng | | | X <sup>&amp;</sup> | x | Х | | | X | X | | | | | | Х | X | X | x | х | X@ |
| 3 | Proced<br>ure<br>(DMR) | Max is 21 days from Baselin e Visit | | | | | | | | | | х | х | Х | | | ¥ | | | | Х | X@ |
| 4 | Day 7<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | х | Х | X@ |
| 5 | Day 14<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | Х | х | X@ |
| 6 | Week 4<br>(28<br>Day) | +/- 7<br>days | | | х | | х | | | | | | | | | х | х | | | Х | х | х |
| 7 | Week 8<br>Call<br>(56<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | Х | | | х | Х | Х |



| 8 | Week<br>12<br>(84<br>Day) | +/- 7<br>days | х | х | | х | х | | | х | х | х | х | Х | х | х |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 9 | Week<br>15 Call<br>(105<br>Day) | +/- 2<br>days | | | | | | | | | Х | | | Х | x | x |
| 10 | Week<br>18<br>(126<br>Day) | +/- 7<br>days | х | х | | | | | | | х | | | Х | х | х |
| 11 | Week<br>21 Call<br>(147<br>Day) | +/- 2<br>days | | | | | | | | | x | | | Х | x | x |
| 12 | Week<br>24<br>(168<br>Day) | +/- 7<br>days | х | х | х | х | | X# | х | | х | х | х | Х | х | х |
| 13 | Week<br>30 Call<br>(210<br>Day) | +/-<br>2days | | | | | | | | | x | | | Х | x | x |
| 14 | Week<br>36<br>(252<br>Day) | + 7<br>days | X | X | | | | | | | X | | | Х | X | x |
| 15 | Week<br>42 Call<br>(294<br>Day) | +/- 2<br>days | | | | | | | | | х | | | X | х | x |
| 16 | Week<br>48<br>(336 | + 7<br>days | Х | х | | х | | | | | | Х | Х | Х | Х | Х |





| | _ | <br> |
|------|---|------|
| Dav) | | |
| Duy, | | |

& for the purpose of eligibility, Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic), for other Blood Pressure assessments it will be measured in a sitting position in duplicate (in same arm) after 15 min of rest

\*Provide diary & glucose meter to the subject

@Subjects using SU will be asked to adjust their SU intake based on section 5.3.1

#A follow up endoscopic evaluation to visually examine the treatment site and adjacent tissues will be conducted after unblinding and within 7 days of visit 12 / week 24

¥The 14-day post procedure diet reviewed with the subject

\*\*Lifestyle Counseling discussions during phone calls at Day 7 & 14 are conducted by the study coordinator in the form of reminders for the subjects and do not need to be conducted by a member of the nutrition staff

Note: Subjects randomized to DMR who do not receive any ablations during the DMR procedure will be followed for safety through the Week 4 visit and then discontinued from the study.

**Table 2: Schedule of Events—Sham Cases** 

| Vis<br>it# | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History &<br>Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pylori Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | Sham / Crossover DMR Procedure | Biopsy | Blinding Assessment | Lífestyle Counseling | SF-36 Quality of Life Questionnaire | PROMIS® Patient Reported<br>Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Diary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Screeni<br>ng<br>(Pre<br>Run-In) | | х | X& | | | x | x | х | | | | | | | | X | | | * | х | x |
| 2 | Baselin<br>e<br>(Post<br>Run-In) | Visit to<br>occur<br>4-6<br>weeks<br>after<br>Screeni | | | X <sup>&amp;</sup> | х | Х | | | Х | х | | | | | | Х | Х | Х | х | х | X@ |



| Vis<br>it# | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History &.<br>Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pylori Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | Sham / Crossover DMR Procedure | Biopsy | Blinding Assessment | Lifestyle Counseling | SF-36 Quality of Life Questionnaire | PROMIS® Patient Reported<br>Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Diary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | ng | | | | | | | | | | | | | | | | | | | | |
| 3 | Proced<br>ure<br>(DMR) | Max is<br>21 days<br>from<br>Baselin<br>e Visit | | | | | | | | | | Х | Х | Х | | | ¥ | | | | Х | X@ |
| 4 | Day 7<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | x | Х | X@ |
| 5 | 14 Day<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | х | X | X@ |
| 6 | Week 4<br>(28<br>Day) | +/- 7<br>days | | | Х | | х | | | | | | | | | Х | х | | | Х | Х | Х |
| 7 | Week 8<br>Call<br>(56<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | Х | | | х | Х | х |
| 8 | Week<br>12<br>(84<br>Day) | +/- 7<br>days | | | x | | х | | | x | х | | | | | х | х | х | х | Х | x | х |
| 9 | Week<br>15 Call<br>(105<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | х | | | Х | Х | х |
| 10 | Week | +/- 7 | | | Х | | Х | | | | | | | | | | Х | | | Х | Х | х |





| Vis<br>it# | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History &<br>Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pylori Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | Sham / Crossover DIMR Procedure | Biopsy | Blinding Assessment | Lifestyle Counseling | SF-36 Quality of Life Questionnaire | PROMIS® Patient Reported<br>Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Diary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 18<br>(126<br>Day) | days | | | | | | | | | | | | | | | | | | | | |
| 11 | Week<br>21 Call<br>(147<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | x | | | х | X | x |
| 12 | Week<br>24<br>(168<br>Day) | +/- 7<br>days | | | х | | х | | х | х | | | | | | | х | х | х | х | х | х |
| 3C | Crossov<br>er to<br>DMR | Within<br>21 days<br>from<br>Week<br>24 | | | | | | | | | | Х | | Х | | | ¥ | | | | Х | х |
| 4C | Crossov<br>er<br>Day 7<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | х | Х | х |
| 5C | Crossov<br>er<br>Day 14<br>Call | +/- 2<br>days | | | | | | | | | | | | | | | ** | | | х | Х | х |
| 6C | Crossov<br>er<br>Week 4<br>(28<br>Day) | +/- 7<br>days | | | х | | х | | | | | | | | | | х | | | х | х | х |



| Vis<br>it# | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History & Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pylori Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | Sham / Crossover DMR Procedure | Biopsy | Blinding Assessment | Lifestyle Counseling | SF-36 Quality of Life Questionnaire | PROMIS® Patient Reported<br>Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Diary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>7</b> C | Crossov<br>er<br>Week 8<br>Call<br>(56<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | х | | | х | х | х |
| 8C | Crossov<br>er<br>Week<br>12<br>(84<br>Day) | +/- 7<br>days | | | х | | х | | | х | х | | | | | | х | х | х | х | х | х |
| 90 | Crossov<br>er<br>Week<br>15 Call<br>(105<br>Day) | +/- 2<br>days | | | | | | | | | | | | | | | х | | | Х | х | х |
| 10<br>C | Crossov<br>er<br>Week<br>18<br>(126<br>Day) | +/- 7<br>days | | | х | | Х | | | | | | | | | | х | | | Х | х | х |
| 11<br>C | Crossov<br>er<br>Week<br>21 Call<br>(147 | +/- 2<br>days | | | | | | | | | | | | | | | Х | | | х | Х | х |



| Vis<br>it# | Visit | Visit Window /<br>Intervention | Informed<br>Consent | History &<br>Full PE | Body Weight & Targeted PE | Pregnancy Test<br>(if applicable) | Blood Analysis | H.pylori Test | ECG | Renal Function | MRE | Endoscopic Evaluation | Subject Randomization &<br>Enrollment | Sham / Crossover DMR Procedure | Biopsy | Blinding Assessment | Lifestyle Counseling | SF-36 Quality of Life Questionnaire | PROMIS® Patient Reported Outcome | Self-Monitoring<br>Blood Glucose/ Glycemia Dlary | Adverse Events | Medication Use® |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day) | | | | | | | | | | | | | | | | | | | | | |
| 12<br>C | Crossov<br>er<br>Week<br>24<br>(168<br>Day) | +/- 7<br>days | | | х | | Х | | Х | х | | | | | | | | Х | Х | Х | х | х |

& for the purpose of eligibility, Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic), for other Blood Pressure assessments it will be measured in a sitting position in duplicate (in same arm) after 15 min of rest

@Subjects using SU will be asked to adjust their SU intake based on section 5.3.1

¥The 14-day post procedure diet reviewed with the subject

\*\*Lifestyle Intervention discussions during phone calls at Day 7 & 14 are conducted by the study coordinator in the form of reminders for the subjects and do not need to be conducted by a member of the nutrition staff

Note: Subjects randomized to Sham who crossover to DMR but do not receive any ablations during the DMR procedure will be followed through the 4 week post crossover visit and then discontinued from the study.

Note: Subjects that choose not to crossover from Sham to DMR will be discontinued from the study and the End of Study CRFs will be completed.

<sup>\*</sup>Provide diary & glucose meter to the subject





#### 4. Statistical Analysis and Reporting

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), median, quartiles, interquartile range (IQR) minimum, and maximum. 95% confidence interval of the mean will be presented where appropriate for efficacy analyses.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment group, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population with non-missing data at each visit.

The minimum and maximum will be reported with the same degree of precision (i.e., the same number of decimal places) as the observed data. Measures of location (mean, quartiles, IQR, and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified and with the following exceptions: a percentage of 0% will not be displayed (i.e., only the count of 0 will be displayed), and a percentage of 100% will be displayed with 0 decimal places.

95% confidence intervals (CIs) will be presented where applicable and will be reported to 1 decimal place. Confidence intervals that cannot be obtained will be displayed as "Not est."

While this protocol does specify primary and safety endpoints, these are not meant to define subject and study success. Instead, the results of this evaluation will be used to establish the safety and efficacy profile of the DMR procedure and to evaluate the effect size for powering future clinical investigations. No *P* values will be reported. More details can be found in Section 

#### 4.2. Interim Analysis and Data Monitoring

It is anticipated that there will be two unblinded deliveries of the data.

1. Week 24 Primary Analysis: The first analysis will occur when all subjects have completed their participation in the randomized treatment phase by either reaching the Week 24 primary endpoint or discontinuing from the study and the data through Week 24 have been frozen. Data through Week 24 will be entered, cleaned, and monitored, and decisions regarding the evaluability of all subject data for inclusion in the primary statistical analysis will be made prior to freezing the data. Other data in the database will





continue to be entered and queried as per normal study conduct. Adverse events (AEs) and concomitant medications that were ongoing at the time of the primary analysis will be unfrozen so the outcomes can be entered for the final analysis.

2. Final Analysis: The second and final analysis will occur when all subjects have completed their participation in the study by either reaching the Week 48 conclusion of the study, or discontinuing, and after the full database has been locked.

Section 13 will delineate which tables, listings, and figures will be provided at each analysis.

#### 4.2.1. Clinical Events Committee

A clinical events committee (CEC) will be established to review important safety AEs reported by trial investigators to determine whether the adjudication of severity and relatedness meets protocol-specified criteria.

Information reviewed on each death, SAE, UADE, or AE of Special Interest (AESI) may include laboratory, pathology and/or imaging data, autopsy reports, physical descriptions, and any other data deemed relevant. The CEC will be masked to the assigned treatment group when performing their assessments. The importance of the CEC is in assessing investigator attribution of causality to the randomized treatment (DMR or Sham) in instances when severity or causality assessments may be deemed subjective and/or require the application of a complex definition.

The CEC will schedule meetings at the following milestones/time points: after the first six (6) subjects, the second set of 6 subjects (total of 12 subjects), and the third set of 6 subjects (total of 18 subjects) have completed visit 6. To allow for adjudication of events following the DMR procedure for Sham subjects who participated in the crossover study, an additional meeting will be scheduled after all crossover Sham subjects have completed visit 6c, Week 4 post procedure. In addition, two other meetings will be scheduled after all DMR subjects complete visit 12, post DMR endoscopic evaluation and biopsy, and Visit 14, 12 weeks post biopsy.

#### **4.2.2. Data Monitoring Committee**

A Data Monitoring Committee (DMC) will be established to conduct reviews of subject safety. It is expected that at least 6 such DMC reviews will occur during the study and they will follow the schedule for the CEC meetings. The DMC reviews will monitor for issues that may justify modifying, suspending, or terminating the study. Only events that have been adjudicated will be used in the DMC safety assessments to guide the DMC decision regarding study continuation. The CEC will not share responsibility with DMC for evaluating interim comparisons; however, their assessments (with results incorporated into the database in a timely manner) will help to ensure that the data reviewed by DMC are as accurate and free of bias as possible.

The sponsor may request additional reviews, e.g., should any other findings/issues pertaining to safety or efficacy emerge requiring DMC review. Details of the operation of the DMC were developed in conjunction with the members of the DMC and can be found in the charter.

The unblinded analysis will be performed by the person responsible for the primary analysis of this study. The DMC listings will not be seen by anyone except the DMC and the performing statistician.





Since there will be no formal hypothesis testing in the summary tables presented in the DMC reports, there will be no statistical penalty.

#### 5. Analysis Populations

The following analysis populations are planned for this study:

- **Study Population**: The study population includes all subjects consented at the site. Within this population there are Screened, Medication Run-In, Intent-to-Treat, As-Treated and Safety populations.
- **Screened Population**: The Screened population includes all subjects who complete Visit 1.
- **Medication Run-In Population:** The Medication Run-In population includes all subjects who entered the Run-In Phase.
- Intent-To-Treat Population (ITT): The ITT population includes all subjects who were randomized after the Medication Run-In phase. This is the secondary analysis population for efficacy. Subjects will be analyzed under the treatment to which they were randomized.
- **As-Treated (AT) Population:** The AT population includes a subset of ITT subjects who received at least one ablation or underwent the randomized Sham procedure. This is the primary population for efficacy. Subjects will be analyzed under the treatment received.
- Week 24 Per Protocol Population: The PP population includes all subjects in the AT population who did not have any major protocol deviations that could affect the assessment of efficacy and had their Week 24 study visit within the protocol-specified window. Subjects will be analyzed under the treatment received.
- Safety Population: The Safety population includes all subjects in whom Sham or DMR procedure was attempted. Subjects will be analyzed according to the treatment received. The Safety population will be further divided into the following 3 sets based on weeks of follow up:
  - Safety population through 24 weeks post-randomization, by treatment received at the start of study
  - Safety population through 24 weeks post-DMR for both treatment groups; this will include the first 24 weeks of the study for subjects receiving DMR from the start of the study and weeks 24-48 post crossover for subjects switching from Sham to DMR. Results will be presented separately for subjects originally receiving DMR, for subjects originally receiving Sham and receiving DMR at week 24, and for all subjects combined receiving DMR at start of the study or at Week 24.
  - Safety population through 48 weeks post-DMR; this will include the 48 weeks of the study for subjects receiving DMR from the start of the study. Results will be presented separately for the first 24 weeks and for Weeks 24-48





The above 3 sets within the Safety population will be identified by period in the summary tables. Period will be categorized as Baseline – Week 24, Week 24 – Week 48, and Baseline – Week 48.

The Baseline – Week 24 period will include the following treatment group columns: DMR, Sham, crossover DMR, and combined DMR. The DMR and Sham treatment group columns will represent the treatment received at the start of the study while the crossover DMR treatment group column will represent the initial Sham recipients who cross over and receive DMR. The combined DMR treatment group column will include all subjects who receive DMR at the start of the study or once they cross over at Week 24.

The Week 24 – Week 48 period will include one column for DMR treatment group, this includes subjects who received DMR at the start of the study.

The Baseline – Week 48 period will also include one column for all subjects overall.

#### 6. General Issues for Statistical Analysis

#### **6.1.** Statistical Definitions and Algorithms

#### 6.1.1. Baseline

The last observation recorded prior to the attempted treatment with index procedure will be used as the baseline observation for all calculations of change from baseline.

#### **6.1.2.** Adjustments for Covariates

Not applicable.

#### **6.1.3.** Multiple Comparisons

No adjustments will be made for multiple comparisons for other endpoints.

#### 6.1.4. Handling of Dropouts or Missing Data

Subjects who withdraw or are withdrawn during screening will be replaced. Subjects who have received the DMR or Sham procedure will be encouraged to complete the end of study procedures.

No imputation will be made for missing data, given the nature of the pilot study. Analyses will be performed using only available data.

#### 6.1.5. Analysis Visit Windows

Visits will be analyzed as scheduled. If a scheduled visit is missing, and an unscheduled/repeated visit exists, the unscheduled/repeated visit will be used in its place; otherwise unscheduled/repeated visits will not be used in the summaries but will be listed.



#### 6.1.6. Pooling of Sites

Not applicable.

#### **6.1.7.** Derived Variables

- **PROMIS**® **Gastrointestinal Nausea and Vomiting Total Score** = sum of the 4 individual items, with a range of 0 to 20, where higher scores indicate worse and more frequent nausea and vomiting. If an individual item is missing, the total score will be set to missing.
- **PROMIS**® **Gastrointestinal Gas and Bloating Total Score** = sum of the 13 individual items, with a range of 0 to 65, where higher scores indicate worse and more frequent gas and bloating. If an individual item is missing, the total score will be set to missing.
- **PROMIS**® **Gastrointestinal Diarrhea Total Score** = sum of the 6 individual items, with a range of 0 to 30, where higher scores indicate worse and more frequent diarrhea. If an individual item is missing, the total score will be set to missing.
- **PROMIS**® **Belly Pain Total Score** = sum of the 5 individual items, with a range of 0 to 25, where higher scores indicate worse and more frequent belly pain. If an individual item is missing, the total score will be set to missing.
- SF-36 Scale Scores<sup>4</sup> = First, precoded numeric values (codelist values) are recoded per the scoring key given in Table 3 where each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Higher scores indicate better quality of life. Second, items in the same scale are averaged together to create the 8 scale scores. Table 4 lists the items averaged together to create each scale. Individual items that are missing are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the subject answered.

**Table 3: Recoding SF-36 Items** 

| SF-36 Item numbers | Change original response category * | To recoded value of: |
|---|---|---|
| 1, 2, 20, 22, 34, 36 | 1 → | 100 |
| | $2 \rightarrow$ | 75 |
| | $3 \rightarrow$ | 50 |
| | $4 \rightarrow$ | 25 |
| | $5 \rightarrow$ | 0 |





| 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 | 1 → | 0 |
|---------------------------------|-----------------|-----|
| 3, 4, 3, 0, 7, 6, 7, 10, 11, 12 | 1 / | |
| | $2 \rightarrow$ | 50 |
| | 3 → | 100 |
| 13, 14, 15, 16, 17, 18, 19 | 1 → | 0 |
| | $2 \rightarrow$ | 100 |
| 21, 23, 26, 27, 30 | 1 → | 100 |
| | $2 \rightarrow$ | 80 |
| | 3 → | 60 |
| | 4 → | 40 |
| | 5 → | 20 |
| | 6 → | 0 |
| 24, 25, 28, 29, 31 | 1 → | 0 |
| | $2 \rightarrow$ | 20 |
| | 3 → | 40 |
| | 4 → | 60 |
| | 5 → | 80 |
| | 6 → | 100 |
| 32, 33, 35 | 1 → | 0 |
| | $2 \rightarrow$ | 25 |
| | 3 → | 50 |
| | 4 → | 75 |
| | 5 → | 100 |



\* Precoded response choices (codelist values) as printed in the SF-36 case report form (CRF).

**Table 4: Averaging Items to SF-36 Scales** 

| Scale | Number of items | After recoding per Table 3, average the following items |
|---|---|---|
| Physical functioning | 10 | 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 |
| Role limitations due to physical health | 4 | 13, 14, 15, 16 |
| Role limitations due to emotional problems | 3 | 17, 18, 19 |
| Energy/fatigue | 4 | 23, 27, 29, 31 |
| Emotional well-being | 5 | 24, 25, 26, 28, 30 |
| Social functioning | 2 | 20, 32 |
| Pain | 2 | 21, 22 |
| General health | 5 | 1, 33, 34, 35, 36 |

- Change from baseline = value at current time point value at baseline
- Percent change from baseline =  $\left(\frac{Change\ from\ baseline\ value}{value\ at\ baseline}\right) * 100$
- **TEAE** = any adverse event with an onset date/time or worsening after index procedure.
- **BMI** =

$$\frac{\textit{weight (kg)}}{\textit{height (cm)}} * \frac{\textit{height (cm)}}{100}$$

- Follow-up time: date of last study visit date of index procedure + 1
- **Duration of diabetes diagnosis:** date of index procedure onset date of first Type 2 diabetes record entered on the medical and diabetic history case report form + 1





#### 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

Adverse events will be coded using the MedDRA version 22.0 thesaurus. Prior and concomitant medications will be coded using the World Health Organization-Drug Dictionary Enhanced (WHO-DDE) (version March 2019) dictionary.

A device- related or procedure-related AE is any AE with a relationship to the study device or procedure of possibly related, probably related, or definitely related.

If partial AE or medication dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows:

For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - If the year matches the year of index procedure date and the end date (if present) is after index procedure date, then impute as the month and day of the index procedure date.
  - o Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the index procedure date, then impute as the day of the index procedure date.
  - o Otherwise, assign 01.

For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - o Otherwise, assign 31 December.



- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

If partial times occur, the convention is as follows:

- if the missing time occurs on the day of the index procedure and both the hour and minute are missing then the time assigned is the time of the index procedure, otherwise if both the hour and minute are missing and the date is not the date of index procedure the time assigned is 12:00;
- if the date is the same as the date of the index procedure and
  - o only hour is missing the hour assigned is 12 or the hour of index procedure, whichever is later;
  - o only the minute is missing the minute assigned is 30 or the minute of index procedure, whichever is later;
- Otherwise if the date is not the same as the date of the index procedure, the hour assigned is 12 if the hour is missing and the minute assigned is 30 if the minute is missing.

#### 7. Study Subjects and Demographics

#### 7.1. Disposition of Subjects and Withdrawals

Disposition will include tabulations of the number of subjects randomized into each treatment group, the number of subjects who received treatment (for subjects randomized to the Sham, that will include subjects who received Sham as well as subjects who received DMR at Week 24), tabulated reasons for discontinuation from the study, and number of subjects in each analysis population. Additionally, summary statistics of follow-up time will be provided. The derivation of follow-up time is provided in Section 6.1.7. The number of subjects completing each follow up visit will also be tabulated.

These summaries will be based on the ITT population.

Inclusion criteria not met and exclusion criteria met and reasons for screen failures will be listed.

#### 7.2. Protocol Violations and Deviations

Protocol deviations (both major and minor), including those due to the impact of COVID-19, as determined by a Sponsor blinded review of the data before database lock and unblinding of the study, may result in the removal of a subject's data from the Week 24 Per Protocol population.

Protocol deviations will be listed. Deviations related to COVID-19 will be listed separately.





Definitions and classifications of major and minor protocol deviations can be found in the study protocol deviation guidance plan.

#### 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, gender, race, ethnicity, height, weight, and body mass index (BMI) will be presented by treatment group using summary statistics or frequencies, as appropriate.

The number and percent of subjects reporting various medical and diabetic histories grouped by MedDRA system organ class and preferred term, will be tabulated. Diabetic history will also be categorized by type of history (diagnosis, symptom, or surgery). The following categories will be used: Type 2 Diabetes, prior therapy, diabetic retinopathy, diabetic nephropathy, diabetic neuropathy, and other. Duration of diabetes diagnosis at baseline will be summarized as part of demographics. The derivation of duration of diabetes diagnosis is provided in Section 6.1.7.

The number of subjects reporting loss of consciousness, admission to hospital, and seizure due to hypoglycemic events in the past year will be tabulated by treatment group. Descriptive statistics on the number of events in the past year will be provided. Targeted hypoglycemic events history will also be listed.

Demographics and baseline characteristics analyses will be conducted for the Medication Run-In, ITT, and AT populations. All other analyses will be conducted for the Safety population only.

#### 7.4. Exposure and Compliance

All subjects will receive the DMR or Sham procedure at the study site under the surveillance of appropriate study personnel and, therefore, no compliance will be calculated. The number of initial Sham recipients who choose to cross-over and receive DMR at Week 24 will be tabulated as part of the disposition summary.

DMR and Sham pre-op and procedure details will be listed separately.

Device use, device malfunctions, and discharge information will be listed.

#### 7.4.1. Endoscopy and Endoscopic Evaluation

On the day of the procedure, subjects will undergo endoscopy with an assessment of the esophagus, stomach, duodenum, and associated structures in order to ensure there are no conditions that would exclude the subject from receiving the index procedure (DMR or Sham). For subjects initially treated with DMR, a follow up endoscopic evaluation to visually examine the treatment site and adjacent tissues will be conducted after all Week 24 Visit assessments are complete and within 7 days of Week 24. During the 24 week follow-up endoscopy, ablation site biopsies will be taken to evaluate the mucosal tissue that has regrown post DMR procedure. For initial Sham subjects who accept the offer to crossover, the endoscopy and DMR procedure will be scheduled within 21 days of the Week 24 Visit.

Endoscopic evaluation results will be tabulated overall. This summary will include presence and grade of esophagitis, duodenum accession and furthest location accessed, abnormalities that would preclude the completion of the DMR procedure, and upper gastrointestinal (GI) conditions. The number of subjects in which the endoscopy procedure was successfully





completed and the number of subjects excluded based on endoscopic findings will also be presented.

Presence and location of ulcers as well as the presence, location, and length of luminal narrowing will be tabulated by treatment group. Visual appearance findings at each location will also be summarized.

All endoscopic evaluation, endoscopy, and duodenal biopsy sample results will be listed.

#### 8. Efficacy Analysis

All efficacy endpoints will be summarized using the AT population as the primary analysis population and repeated on the ITT population. The primary efficacy analysis will also be repeated in the Week 24 Per Protocol population. All efficacy data, regardless of population, will be presented in data listings.

#### 8.1. Primary Efficacy Analysis

The primary efficacy endpoint is the change in HbA1c at Week 24. Descriptive statistics of observed, change from baseline, and percent change from baseline to Week 24 HbA1c values will also be provided by treatment group. 95% CI of the mean will also be presented.

#### 8.2. Secondary Efficacy Analysis

#### 8.2.1. HbA1c Over Time

Descriptive statistics of observed, change from baseline, and percent change from baseline to each study visit through Week 24 HbA1c will also be provided by treatment group and study visit. 95% CI of the mean will also be presented.

The proportion of subjects with an HbA1c improvement from baseline at Week 24 that maintain an HbA1c improvement at Week 48 will be presented for DMR treatment group subjects. An improvement in HbA1c is defined as any value lower than baseline.

Descriptive statistics of the end-of-Run-In-phase HbA1c for all Medication Run-In subjects will also be presented overall.

#### 8.2.2. Fasting Plasma Glucose (FPG)

Descriptive statistics of observed, change from baseline, and percent change from baseline to each study visit through Week 24 FPG will also be provided by treatment group and study visit. 95% CI of the mean will also be presented.

#### 8.2.3. Urine Albumin Creatinine Ratio (UACR)

Descriptive statistics of observed, change from baseline, and percent change from baseline to each study visit through Week 24 UACR will also be provided by treatment group and study visit. 95% CI of the mean will also be presented.



#### 8.2.4. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)

Descriptive statistics of observed, change from baseline, and percent change from baseline to each study visit through Week 24 ALT and AST will also be provided by treatment group and study visit. 95% CI of the mean will also be presented.

#### 8.3. Additional Endpoints of Interest

The above secondary analyses of HbA1c, FPG, UACR, ALT, and AST will also be repeated from baseline through Week 48 for the DMR treatment group by study visit.

For initial Sham recipients, descriptive statistics of observed, change from Week 24 (pre-DMR) to Week 48, and percent change from Week 24 (pre-DMR) to Week 48 will also be displayed for HbA1c and FPG. 95% CI of the mean will be presented.

#### 8.3.1. Short Form (36) Health Survey (SF-36)

Subjects will complete an assessment of health status and quality of life, the SF-36 Questionnaire, at Baseline, Week 12, Week 24 and Week 48. These measures rely upon subject self-reporting. The SF-36 asks 36 questions to measure functional health and well-being from the subject's point of view and taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Derivations for each of the scale scores are described in Section 6.1.7.

Change from baseline to study visit in the physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health scale scores will be summarized by treatment group and study visit.

#### 8.3.2. Patient Reported Outcomes Measurement Information System (PROMIS®)

Subjects will complete the PROMIS® at Baseline, Week 12, Week 24 and Week 48. PROMIS® is a set of person-centered measures that will be used to evaluate and monitor physical health in subjects. For the purposes of this study, the gastrointestinal symptom domains were chosen including nausea/vomiting, gas/bloating, diarrhea, and belly pain. Derivations for each of the total scores are described in Section 6.1.7.

Change from baseline to study visit in the PROMIS® Gastrointestinal Nausea and Vomiting Total Score, Gastrointestinal Gas and Bloating Total Score, Gastrointestinal Diarrhea Total Score, and Belly Pain Total Score will be summarized by treatment group and study visit.

#### 9. Safety and Tolerability Analysis

Safety variables include AEs, SAEs, UADEs, vital sign measurements, weight, physical exam findings, laboratory test results, 12-lead ECG findings, and MRE findings. No formal inferential analyses are planned for the safety endpoints.





#### 9.1. Adverse Events

All AEs that start or worsen after the time of index procedure will be considered TEAEs. Events meeting this definition will be those events that are a change from the subject's baseline conditions, including an increase in frequency or severity (these will be entered as new AEs). For AEs occurring on the date of index procedure, if the time of onset is missing, the AE will be assumed to be treatment emergent.

All AEs, TEAEs, and SAEs will be coded using the MedDRA Version 22.0 or higher coding dictionary. The AE analyses will focus on those that are treatment emergent, however any AEs that are reported after consent has been signed and before initial dosing will included in the listings.

The causal relationship of the AE to the study device and the study procedure is determined by the investigator as Not Related, Possibly Related, Probably Related, or Definitely Related. These can be mapped to Not Related (*Not Related*) and Related (*Possibly Related*, *Probably Related* and *Definitely Related*). Adverse event summaries will be repeated for treatment related TEAEs.

Adverse events severity grades are reported as mild, moderate, or severe.

Summaries of incidence rates (frequencies and percentages) of individual TEAEs will be presented by SOC, PT, period, and treatment group. Period is defined in Section 5. Such summaries will be displayed for all TEAEs, TEAEs by maximum severity, and TEAEs by relationship to device and/or procedure. Incidence of TEAEs during the Medication Run-In phase will also be presented by SOC and PT for the Medication Run-In population.

Each subject will be counted only once within each summation level (SOC and PT). If a subject experiences more than 1 TEAE within each summation level only, the TEAE with the strongest relationship or the maximum severity, as appropriate, will be included in the summaries of relationship and severity. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = definitely related). If a subject has separate AEs with the same SOC/PT with one starting in the double-blind period and the other starting after Week 24, they are counted once within each period.

Incidences will be presented by descending frequency of SOC and PT within SOC, and then alphabetically within PT where the incidence is the same; this is based on overall subjects then alphabetically in case of a tie.

Missing and partially missing AE start and/or stop dates will be imputed, for the purpose of statistical analysis, according to the specifications described in Section 6.1.8.

In the AE data listings, all AEs will be displayed. AEs that are treatment emergent will be flagged.

#### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to withdrawal from the study, by period, treatment group, SOC, and preferred term will be prepared for the





Safety Population. TEAEs leading to withdrawal will also be tabulated by relationship to device and procedure.

A data listing of AEs leading to withdrawal from the study will also be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occur during the study will be listed.

Serious adverse events will be listed and also tabulated by system organ class and preferred term and presented by period and treatment group. SAEs will also be tabulated by relationship to device and procedure.

#### 9.1.3. Other Significant Adverse Events

A review of AEs will be performed prior to database lock and those related to COVID-19 will be flagged separately and summarized by SOC, PT and treatment group.

#### 9.1.3.1. Unanticipated Adverse Device Effects (UADEs)

A summary of incidence rates (frequencies and percentages) of UADEs by period, treatment group, SOC, and preferred term will be prepared for the Safety Population. UADEs will also be tabulated by relationship to device and procedure.

Unanticipated adverse device effects will be flagged in the AE listing.

#### 9.1.3.2. Adverse Events of Special Interest (AESIs)

Adverse events of special interest include the following:

- Hypoglycemia
- Diarrhea
- Abdominal pain
- Nausea
- Vomiting
- Gastrointestinal bleeding
- Unexplained fever

A summary of AESIs by period, treatment group, SOC, and preferred term will be prepared for the Safety Population. All AESIs will be flagged in the AE listing.

Episodes of diarrhea will be recorded both as events and as incidence.

Descriptive statistics on the blood glucose values and duration of episode reported on the hypoglycemia form will be provided as will summaries of treatment and symptoms. Additionally, the incidence and event rates of hypoglycemia will be tabulated by severity of the hypoglycemia: severe hypoglycemic event, defined as hypoglycemia requiring third-party assistance; or any clinically significant hypoglycemic event, defined as self-monitored or laboratory plasma glucose level < 54 mg/dL (3.0 mmol/L); or glucose alert values  $\leq$ 70 mg/dL





(3.9 mmol/L).

All hypoglycemia cases will be listed.

Patient contact regarding hypoglycemia will also be listed as will blood glucose and glycemia diary details. Hyperglycemia rescue data will be listed separately.

#### 9.2. Clinical Laboratory Evaluations

Laboratory test results (complete blood count, blood chemistry, liver panel, pancreatic enzymes, thyroid stimulating hormone [TSH], fasting lipid panel, FPG, HbA1c, fasting C-Peptide, and fasting insulin) will be summarized descriptively by treatment group and study visit as both observed values and change from baseline values. H. Pylori results will only be listed as it is only collected at screening.

The number of subjects with clinical laboratory values below, within, or above normal ranges, by study visit, will be tabulated (shift tables) for each clinical laboratory analyte by period and treatment group.

Laboratory values will be displayed in the data listings, and those that are outside the normal range will be flagged and presented, along with corresponding normal ranges (if available).

A separate listing of abnormal laboratory values, including renal function, will be provided. All study visits within an analyte for a subject will be presented if at least 1 study visit within that analyte has an abnormal result.

Pregnancy test results will be listed separately.

#### 9.3. Vital Signs

Vital signs will be collected at Screening, Baseline, Week 4, Week 12, Week 18, Week 24, Week 36, and Week 48.

Descriptive summaries of observed values and changes from baseline will be calculated for weight (kg), sitting systolic blood pressure (mmHg), sitting diastolic blood pressure (mmHg), and pulse rate (bpm).

Vital signs measurements will also be listed.

#### 9.4. Electrocardiograms

12-Lead electrocardiograms will be obtained at Screening and Week 24.

Descriptive summaries will be presented for ECG measures of PR interval (msec), RR interval (msec), ventricular rate (bpm), QRS interval (msec), uncorrected QT interval (ms), QTcB interval (ms), and investigator interpretation. These summaries will be presented by study visit and treatment group.

12-lead ECG results will also be listed.




### 9.5. Further Safety Evaluations

## 9.5.1. MRI Enterography

Clinically relevant abnormal findings from the central MRE reader will be listed.

## 9.5.2. Lifestyle Counseling and Evaluation

Lifestyle counseling and evaluation data will be listed.

### 9.6. Concomitant Medication

Prior and concomitant medications, coded using World Health Organization drug dictionary (WHO-DDE) (March 2019), will be summarized descriptively by Anatomical Therapeutic Chemical (ATC) classification Level 4 and PT (i.e., ATC classification Level 5), if applicable, and by period and treatment group using counts and percentages.

Prior medications will be presented separately from concomitant medications. The assignment of medications as prior and/or concomitant will be done as follows:

- **Prior medications:** Medications that started before the index procedure will be considered prior medications whether or not they were stopped before the index procedure.
- **Concomitant medications:** Any medications continuing or starting after the index procedure through the end of study will be considered to be concomitant.

If a medication starts prior to the index procedure and continues after the index procedure it will be considered both prior and concomitant. Prior and concomitant medications will also be listed.

### 9.7. Physical Exam

A full physical examination will be performed at Screening to assess the following organ systems: general appearance, cardiovascular, respiratory, lymph nodes, neurological, skin, head, eyes, ears, nose, and throat, extremities, musculoskeletal, genitourinary, funduscopic exam, thyroid palpation, abdominal exam, heart and lung auscultation, deep tendon reflex and sensation (vibration, pinprick) assessment in distal lower extremities. A targeted physical exam will be performed at Baseline Week 4, Week 12, Week 18, Week 24, Week 36, and Week 48 to assess the following systems: funduscopic exam, thyroid palpation, abdominal exam, heart and lung auscultation, deep tendon reflex and sensation (vibration, pinprick) assessment in distal lower extremities.

All physical exam results will be listed by body system and both abnormal and clinically significant results will be flagged.

### 10. Changes from Planned Analysis

The Screened and Medication Run In analysis populations were not defined in the protocol; thus, they are defined in this SAP.





An additional analysis population, the Week 24 Per Protocol population was added, to determine the impact of protocol deviations, especially those that are a result of the COVID-19 pandemic, and out of window visits on primary efficacy results.

Significance testing and statistical modeling will be omitted due to the small sample size. The results of this pilot study will be used to establish the safety and efficacy profile of the DMR procedure and to evaluate the effect size for powering future clinical investigations, therefore no formal comparisons within or between treatment groups will be performed.

## 11. Other Planned Analysis

Not Applicable.





#### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. SF-36 Scoring <a href="https://www.rand.org/health-care/surveys\_tools/mos/36-item-short-form/scoring.html">https://www.rand.org/health-care/surveys\_tools/mos/36-item-short-form/scoring.html</a>

## 13. Tables, Listings, and Figures

All listings, tables, and figures will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (CRF page or listing number).

The following reporting conventions will be adopted for the presentation of study data. These conventions will enhance the review process and help to standardize the presentation with common notations.

## **General Reporting Conventions**

- All tables and data listings will be developed in landscape orientation.
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters should be used in tables and data listings. Special characters, such as nonprintable control characters, printer-specific characters, or font specific characters, will not be used on a table, figure, or data listing.
- Adverse events with missing MedDRA coding will have their system organ class and/or preferred term presented as "Not Coded" in the tables. The "Not Coded" frequencies will be sorted to the end of the tables. This will only be applicable for any deliveries sent before database lock (e.g., for dry runs on blinded data).
- Programming notes may be inserted into the shells, these notes will not appear in the final output.

### **Population Summary Conventions**

- Population sizes may be presented for each classification factor as totals in the column header as (N=xxx), where appropriate.
- All population summaries for categorical variables will include all categories that were planned and for which the subjects may have had a response. Percentages corresponding

Statistical Analysis Plan, Sponsor Fractyl Laboratories Inc. Protocol Number C-40000 PCN Number FRAC8070



to null categories (cells) will be suppressed; however, counts and percentages of missing values may be needed.

- All population summaries for continuous variables will include: N, mean, SD, median, quartiles, IQR, minimum, and maximum. Other summaries (e.g., number missing or 95% CIs) may be used as appropriate.
- See Section 4.1 for specifications for rounding.

## 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number C-40000. The table numbers and page numbers are place holders only and will be determined when the tables are produced.



# Table 5: Demographic Data Summary Tables and Figures

| Number | Population | Title | Unique/Non-<br>Unique | Provide at Topline? |
|---|---|---|---|---|
| Table 14.1.1.1 | ITT | Summary of Subject Disposition and Follow Up<br>Compliance | Unique | |
| Table 14.1.1.2 | | Summary of Analysis Population Eligiblities | Unique | |
| Table 14.1.2.1 | Medication<br>Run-In | Demographics and Baseline Characteristics | Unique | |
| Table 14.1.2.2 | ITT | Demographics and Baseline Characteristics | Non-Unique | |
| Table 14.1.2.3 | AT | Demographics and Baseline Characteristics | Non-Unique | X |
| Table 14.1.3.1 | Safety | Summary of Medical History by SOC, PT, and Treatment | Unique | |
| Table 14.1.3.2 | Safety | Summary of Diabetic History by SOC, PT, and Treatment | Non-Unique | |
| Table 14.1.3.3 | Safety | Summary of Targeted Hypoglycemic Events History by Treatment | Unique | |
| Table 14.1.4 | Safety | Summary of Prior Medications by ATC Class Level 4, PT, and Treatment | Unique | |
| Table 14.1.5.1 | Medication<br>Run-In | Summary of Endoscopic Evaluation | Unique | |
| Table 14.1.5.2 | Safety | Summary of Endoscopy Results | Unique | |

# 13.2. Efficacy Data

# **Table 6: Efficacy Data**

| Number | Population | Title | Unique/Non-<br>Unique | Provide at Topline? |
|---|---|---|---|---|
| Table 14.2.1.1 | AT | Summary of Change from Baseline in HbA1c by Study Visit and Treatment | Unique | X |
| Table 14.2.1.2 | ITT | Summary of Change from Baseline in HbA1c by Study Visit and Treatment | Non-Unique | |
| Table 14.2.1.3 | Week 24 Per<br>Protocol | Summary of Change from Baseline in HbA1c by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.2.1.4 | Medication<br>Run-In | Summary of HbA1c During Medication Run-In | Non-Unique | |
| Table 14.2.1.5 | AT | Summary of Change from Week 24 in HbA1c by Study Visit and Treatment | Non-Unique | |
| Table 14.2.1.6 | ITT | Summary of Change from Week 24 in HbA1c by Study Visit and Treatment | Non-Unique | |



| Number | Population | Title | Unique/Non-<br>Unique | Provide at Topline? |
|---|---|---|---|---|
| Table 14.2.1.7 | AT | Summary of HbA1c Improvement by Study Visit and Treatment | Unique | |
| Table 14.2.1.8 | ITT | Summary of HbA1c Improvement by Study<br>Visit and Treatment | Non-Unique | |
| Table 14.2.1.9 | Week 24 Per<br>Protocol | Summary of HbA1c Improvement by Study<br>Visit and Treatment | Non-Unique | |
| Table 14.2.2.1 | AT | Summary of Change from Baseline in FPG by Study Visit and Treatment | Non-Unique | X |
| Table 14.2.2.2 | ITT | Summary of Change from Baseline in FPG by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.2.2.3 | AT | Summary of Change from Week 24 in FPG by Study Visit and Treatment | Non-Unique | |
| Table 14.2.2.4 | ITT | Summary of Change from Week 24 in FPG by Study Visit and Treatment | Non-Unique | |
| Table 14.2.3.1 | AT | Summary of Change from Baseline in UACR by Study Visit and Treatment | Non-Unique | X |
| Table 14.2.3.2 | ITT | Summary of Change from Baseline in UACR by Study Visit and Treatment | Non-Unique | |
| Table 14.2.4.1 | AT | Summary of Change from Baseline in ALT by<br>Study Visit and Treatment | Non-Unique | X |
| Table 14.2.4.2 | ITT | Summary of Change from Baseline in ALT by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.2.5.1 | AT | Summary of Change from Baseline in AST by<br>Study Visit and Treatment | Non-Unique X | |
| Table 14.2.5.2 | ITT | Summary of Change from Baseline in AST by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.2.6.1 | AT | Summary of Change from Baseline in SF-36<br>Scale Scores by Study Visit and Treatment | Non-Unique | |
| Table 14.2.6.2 | ITT | Summary of Change from Baseline in SF-36<br>Scale Scores by Study Visit and Treatment | Non-Unique | |
| Table 14.2.7.1 | AT | Summary of Change from Baseline in PROMIS<br>Scores by Study Visit and Treatment | Non-Unique | |
| Table 14.2.7.2 | ITT | Summary of Change from Baseline in PROMIS<br>Scores by Study Visit and Treatment | Non-Unique | |

## 13.3. Safety Data

**Table 7: Safety Data** 



| Number | Population | Title | Unique/Non-<br>Unique | Provide at Topline? |
|---|---|---|---|---|
| 14.3.1 Dis | plays of Adv | erse Events | | |
| Table 14.3.1.1 | Safety | Summary of Adverse Events by Treatment | Unique | |
| Table 14.3.1.2 | Safety | Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment | Unique | X |
| Table 14.3.1.3 | Safety | Incidence of Treatment Emergent Adverse Events by<br>Maximum Severity, SOC, PT, and Treatment | Unique | |
| Table 14.3.1.4 | Safety | Incidence of Treatment Emergent Adverse Events by<br>Relationship, SOC, PT, and Treatment | Unique | |
| 1 | 4.3.2 Summa | ary of Deaths, Other Serious and Significant Adverse E | vents | |
| Table 14.3.2.1 | Safety | Incidence of Adverse Events Leading to Withdrawal by SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.2 | Safety | Incidence of Adverse Events Leading to Withdrawal by Relationship, SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.3 | Safety | Incidence of Serious Adverse Events by SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.4 | Safety | Incidence of Serious Adverse Events by Relationship, SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.5 | Safety | Incidence of Unanticipated Adverse Device Effects by SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.6 | Safety | Incidence of Unanticipated Adverse Device Effects by<br>Relationship, SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.7 | Safety | Incidence of Adverse Events of Special Interest by SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.8 | Safety | Incidence of COVID-19 Adverse Events by SOC, PT, and Treatment | Non-Unique | |
| Table 14.3.2.9 | Safety | Summary of Hypoglycemic Events by Treatment | Unique | |
| Table 14.3.2.10 | Safety | Summary of Diarrhea by Treatment | Unique | |
| 14.3.3 Na | arratives of I | Deaths, Other Serious and Certain Other Significant Ad | verse Events | |
| Table 14.3.3.1 | Safety | Listing of Adverse Events Leading to Withdrawal | Unique | |
| Table 14.3.3.2 | Safety | Listing of Serious Adverse Events | Non-Unique | |
| Table 14.3.3.3 | Safety | Listing of Deaths | Non-Unique | |



| Number | Population | Title | Unique/Non-<br>Unique | Provide at Topline? |
|---|---|---|---|---|
| Table 14.3.3.4 | Safety | Listing of Unanticipated Adverse Device Effects | Non-Unique | |
| Table 14.3.3.5 | Safety | Listing of Adverse Events of Special Interest | Non-Unique | |
| 14.3.4 Abı | normal Labo | ratory Value | | |
| 14.3.4.1 | Safety | Listing of Abnormal Laboratory Data | Unique | |
| 14.3.5 Lab | oratory Dat | a Summary Tables | | |
| Table 14.3.5.1.1 | Safety | Summary of Complete Blood Count Laboratory Results by Study Visit and Treatment | Unique | |
| Table 14.3.5.1.2 | Safety | Shift from Baseline in Complete Blood Count<br>Laboratory Results by Study Visit and Treatment | Unique | |
| Table 14.3.5.2.1 | Safety | Summary of Blood Chemistry Laboratory Results by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.3.5.2.2 | Safety | Shift from Baseline in Blood Chemistry Laboratory<br>Results by Study Visit and Treatment | Non-Unique | |
| Table 14.3.5.3.1 | Safety | Summary of Urinalysis Laboratory Results by Study<br>Visit and Treatment | Non-Unique | |
| Table 14.3.5.3.2 | Safety | Shift from Baseline in Urinalysis Laboratory Results by<br>Study Visit and Treatment | Non-Unique | |
| 14.3.6 Oth | er Safety Da | nta Summary Tables | | |
| Table 14.3.6.1.1 | Safety | Summary of Vital Signs by Study Visit and Treatment | Non-Unique | X |
| Table 14.3.6.2.1 | Safety | Summary of 12-Lead Electrocardiogram Results by<br>Study Visit and Treatment | Non-Unique | |
| Table 14.3.6.2.2 | Safety | Summary of 12-Lead Electrocardiogram Interpretation by Study Visit and Treatment | Unique | |
| Table 14.3.6.3.1 | Safety | Summary of Concomitant Medications by ATC Class<br>Level 4, PT, and Treatment | Unique | |





## 13.4. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number C-40000.

In general, one listing will be produced per CRF domain. All listings will be sorted by treatment, site, and subject number. Listings will also be sorted by date and time of assessment, if applicable. Screen failures will only be presented in Listings 16.2.2.1 and 16.2.3.

All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (e.g., repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 8: Planned Listings** 

| Number | Dataset | Title / Summary | Unique/Non-<br>Unique |
|---|---|---|---|
| 16.2.1 Subject D | iscontinuati | ions/Completions | |
| Listing 16.2.1 | All<br>Subjects | Subject Disposition | Unique |
| 16.2.2 Protocol l | Deviations | | |
| Listing 16.2.2.1 | All<br>Subjects | Inclusion and Exclusion Criteria Not Met | Unique |
| Listing 16.2.2.2.1 | All<br>Subjects | Protocol Deviations | Unique |
| Listing 16.2.2.2.2 | All<br>Subjects | COVID-19 Protocol Deviations | Non-nique |
| 16.2.3 Subjects l | Excluded fro | om the Efficacy Analyses | |
| Listing 16.2.3 | All<br>Subjects | Analysis Populations | Unique |
| 16.2.4 Demogra | phic Data aı | nd Other Baseline Characteristics | |
| Listing 16.2.4.1 | All<br>Subjects | Demographics and Baseline Characteristics | Unique |
| Listing 16.2.4.2.1 | All<br>Subjects | Diabetic History | Unique |
| Listing 16.2.4.2.2 | All<br>Subjects | Medical History | Unique |
| Listing 16.2.4.2.3 | All<br>Subjects | Targeted Hypoglycemic Events History | Unique |
| 16.2.5 Complian | ce and/or D | rug Concentration Data | |



| Number | Dataset | Title / Summary | Unique/Non-<br>Unique |
|---|---|---|---|
| Listing 16.2.5.1.1 | All<br>Subjects | DMR Procedure Pre-Op | Unique |
| Listing 16.2.5.1.2 | All<br>Subjects | DMR Procedure Lift and Ablation Details | Unique |
| Listing 16.2.5.2.1 | All<br>Subjects | Sham Procedure Pre-Op | Unique |
| Listing 16.2.5.2.2 | All<br>Subjects | Sham Procedure Details | Unique |
| Listing 16.2.5.3.1 | All<br>Subjects | Device Use Summary | Unique |
| Listing 16.2.5.3.2 | All<br>Subjects | Device Malfunction | Unique |
| Listing 16.2.5.4.1 | All<br>Subjects | Endoscopic Evaluation | Unique |
| Listing 16.2.5.4.2 | All<br>Subjects | Endoscopy | Unique |
| Listing 16.2.5.4.3 | All<br>Subjects | Biopsy | Unique |
| Listing 16.2.5.5.1 | All<br>Subjects | Discharge Information | Unique |
| 16.2.6 Individua | l Efficacy Re | esponse Data | |
| Listing 16.2.6.1 | All<br>Subjects | HbA1c | Unique |
| Listing 16.2.6.2 | All<br>Subjects | Fasting Plasma Glucose (FPG) | Non-Unique |
| Listing 16.2.6.3 | All<br>Subjects | Urine Albumin Creatinine Ratio (UACR) | Non-Unique |
| Listing 16.2.6.4 | All<br>Subjects | Alanine Aminotransferase (ALT) | Non-Unique |
| Listing 16.2.6.5 | All<br>Subjects | Aspartate Aminotransferase (AST) | Non-Unique |
| Listing 16.2.6.6 | All<br>Subjects | SF-36 Quality of Life Questionnaire | Unique |
| Listing 16.2.6.7 | All<br>Subjects | PROMIS Scores | Unique |
| 16.2.7 Adverse E | Event Listing | s (by Subject) | |
| Listing 16.2.7.1 | All<br>Subjects | Adverse Events | Non-Unique |



| Number | Dataset | Title / Summary | Unique/Non-<br>Unique |
|---|---|---|---|
| Listing 16.2.7.2 | All<br>Subjects | Hypoglycemia Form | Non-Unique |
| 16.2.8 Laborator<br>Subject) | ry Values an | d Other Clinical Observations and Measurements (by | |
| Listing 16.2.8.1.1 | All<br>Subjects | Laboratory Data: Complete Blood Count | Non-Unique |
| Listing 16.2.8.1.2 | All<br>Subjects | Laboratory Data: Blood Chemistry | Non-Unique |
| Listing 16.2.8.1.3 | All<br>Subjects | Laboratory Data: Urinalysis | Non-Unique |
| Listing 16.2.8.1.4 | All<br>Subjects | Urine Pregnancy Test | Unique |
| Listing 16.2.8.1.5 | All<br>Subjects | Self Monitoring Blood Glucose and Glycemia Diary | Unique |
| Listing 16.2.8.2.1 | All<br>Subjects | Vital Signs | Unique |
| Listing 16.2.8.3 | All<br>Subjects | 12-Lead Electrocardiogram (ECG) Results | Unique |
| Listing 16.2.8.4 | All<br>Subjects | MRI Enterography (MRE) | Unique |
| Listing 16.2.8.5.1 | All<br>Subjects | Lifestyle Counseling | Unique |
| Listing 16.2.8.5.2 | All<br>Subjects | Lifestyle Evaluation | Unique |
| Listing 16.2.8.6 | All<br>Subjects | Prior and Concomitant Medications | Unique |
| Listing 16.2.8.7.1 | All<br>Subjects | Physical Examination | Unique |
| Listing 16.2.8.7.2 | All<br>Subjects | Targeted Physical Examination | Non-Unique |
| Listing 16.2.8.8.1 | All<br>Subjects | Patient Contact | Unique |
| Listing 16.2.8.8.2 | All<br>Subjects | Day 7 Telephone Contact | Unique |
| Listing 16.2.8.8.3 | All<br>Subjects | Day 14 Telephone Contact | Unique |
| Listing 16.2.8.8.4 | All<br>Subjects | Telephone Contact | Unique |





| Number | Dataset | Title / Summary | Unique/Non-<br>Unique |
|---|---|---|---|
| Listing 16.2.8.8.5 | All<br>Subjects | Follow Up Office Visit | Unique |





## 14. Tables, Listings, and Listing Shells

# 14.1. Standard Layout for all Tables, Listings, and Figures

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each TLF shell.





# Figure 1: Standardized Layout

| Fractyl Laboratories | Page xx of xx |
|---|---|
| Protocol: C-40000 | Version |
| <table, figure="" listing,=""> xx.x.x</table,> | |
| <title figure="" listing,="" of="" or="" table,="">&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If directly Applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 1 &lt;if applicable&gt; Recommendation is to keep footnotes to a minimum&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 2 &lt;if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n &lt;if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n+1 &lt;pgm path and name&gt;, &lt;date&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |





## 14.2. Planned Table Shells

See Figure 2 below.



Figure 2: Planned Table Shells

Table 14.1.1.1 Summary of Subject Disposition and Follow-up Compliance by Treatment **ITT** Population

| | DMR | Sham | Overall |
|--------------------------------|--------------|--------------|--------------|
| Status | (N=XX) | (N=XX) | (N=XX) |
| Completed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Early Termination | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reason for Early Termination: | | | |
| Adverse Event | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lost to Follow-up | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Physician Decision | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Protocol Violation | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Study Terminated by Sponsor | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Withdrawal by Subject | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Crossed Over to DMR at Week 24 | | XX (XX.X%) | XX (XX.X%) |
| Completed Week 4 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Week 12 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Week 18 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Week 24 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Week 36 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Completed Week 48 Visit | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Follow-up Time (days) | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range; ITT = intent to treat.

Note: Percentages are n/Number of subjects in the ITT population\*100. Subjects are summarized by randomized treatment and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Follow-up time is derived as the date of last study visit – date of index procedure + 1. IQR = Q3 – Q1.

SOURCE: Listing 16.2.1

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.1.1.2
Summary of Analysis Population Eligibilities by Treatment

| Status | DMR<br>(N=XX) | Sham<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Study Population [1] | | | XX |
| Screened Population [2] | | | XX |
| Medication Run-In Population [3] | | | XX |
| TT Population [4] | XX | XX | XX |
| As-Treated Population [5] | XX | XX | XX |
| Week 24 Per-Protocol Population [6] | XX | XX | XX |
| Safety Population [7] | XX | XX | XX |

Abbreviations: DMR = duodenal mucosal resurfacing; ITT = intent to treat; PP = per-protocol.

Note: Subjects are summarized by randomized treatment and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Follow-up time is derived as the date of last study visit – date of index procedure + 1.

- [1] The Study Population includes all subjects consented at the site.
- [2] The Screened population includes all subjects who completed Visit 1.
- [3] The Medication Run-In population includes all subjects who entered the Run-In Phase.
- [4] The ITT Population includes all subjects who were randomized after the Medication Run-In phase.
- [5] The As-Treated Population is a subset of ITT subjects who received at least one ablation or underwent the randomized Sham procedure.
- [6] The PP population includes all subjects in the AT population who did not have any major protocol deviations that could affect the assessment of efficacy and had their Week 24 study visit within the protocol-specified window.
- [7] The Safety Population includes all subjects in whom Sham or DMR was attempted.

SOURCE: Listing 16.2.1





# Table 14.1.2.1 Summary of Demographics and Baseline Characteristics Medication Run-In Population

| Variable Statistic or Catagonia | Overall (N-VV) |
|----------------------------------------------|--------------------------|
| Statistic or Category | (N=XX) |
| Age (years) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |
| Sex | |
| Male | XX (XX.X%) |
| Female | XX (XX.X%) |
| Child-bearing Age? [1] | XX (XX.X%) |
| Edhariaita. | |
| Ethnicity Hispania or Latina | VV (VV V0/ ) |
| Hispanic or Latino<br>Not Hispanic or Latino | XX (XX.X%)<br>XX (XX.X%) |
| Not Reported | XX (XX.X%)<br>XX (XX.X%) |
| Unknown | XX (XX.X%) |
| CHARLEM | 70((701.7770) |
| Race | |
| American-Indian or Alaska Native | XX (XX.X%) |
| Asian | XX (XX.X%) |
| Black or African-American | XX (XX.X%) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X%) |
| White | XX (XX.X%) |
| More than One Race | XX (XX.X%) |
| Race not Provided | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Medication Run-In Population\*100. Subjects are summarized overall. IQR = Q3 – Q1.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety Population.

SOURCE: Listing 16.2.4.1





# Table 14.1.2.1 (cont.) Summary of Demographics and Baseline Characteristics Medication Run-In Population

| Variable | Overall |
|-------------------------|--------------|
| Statistic or Category | (N=XX) |
| Height (cm) | |
| n ' | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |
| Weight (kg) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |
| | 74,75 |
| Body Mass Index (kg/m²) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Medication Run-In Population\*100. Subjects are summarized overall. Duration of Type 2 Diabetes diagnosis is derived as the date of index procedure — onset date of first Type 2 diabetes record entered on the medical and diabetic history case report form + 1. IQR = Q3 - Q1.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety Population.

SOURCE: Listing 16.2.4.1





# Table 14.1.2.1 (cont.) Summary of Demographics and Baseline Characteristics Medication Run-In Population

| Variable | Overall |
|---------------------------------------|--------------|
| Statistic or Category | (N=XX) |
| HbA1c (mmol/mol) | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | xx.x |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |
| Duration of Type 2 Diabetes Diagnosis | |
| n | XX |
| Mean (SD) | XX.X (XX.XX) |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| IQR | XX.X |
| Min, Max | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Medication Run-In Population\*100. Subjects are summarized overall. Duration of Type 2 Diabetes diagnosis is derived as the date of index procedure – onset date of first Type 2 diabetes record entered on the medical and diabetic history case report form + 1. IQR = Q3 - Q1.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Safety Population.

SOURCE: Listing 16.2.4.1





#### Table 14.1.2.2 Summary of Demographics and Baseline Characteristics by Treatment ITT Population

#### Same shell as Table 14.1.2.1

**Programing note:** Add ITT (Intent-to-Treat) to abbreviations. Update footnote to read "Note: Percentages are n/Number of subjects in the ITT Population\*100. Subjects are summarized by randomized treatment and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Include two columns for DMR and Sham and display them before the Overall column, as shown below.

| Variable | DMR | Sham | Overall |
|-----------------------|--------|--------|---------|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |

# Table 14.1.2.3 Summary of Demographics and Baseline Characteristics by Treatment AT Population

#### Same shell as Table 14.1.2.1

**Programing note:** Add AT (As-Treated) to abbreviations. Update footnote to read "Note: Percentages are n/Number of subjects in the AT Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Include two columns for DMR and Sham and display them before the Overall column, as shown below.

| Variable | DMR | Sham | Overall |
|-----------------------|--------|--------|---------|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |





Table 14.1.3.1 Summary of Medical History by SOC, PT, and Treatment Safety Population

| System Organ Class<br>Preferred Term | DMR<br>(N=XX) | Sham<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Subjects with at least 1 Recorded Non-DiabeticMedical History | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; PT = Preferred Term; SOC = System Organ Class. Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Medical histories were coded using MedDRA version 22.0. Subjects were counted once for each system organ class (SOC) and once for each preferred term (PT). Medical history terms are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.4.2.2

Programming note: Ensure proper MedDRA version is displayed in footnote.





Table 14.1.3.2 Summary of Diabetic History by SOC, PT, and Treatment Safety Population

| System Organ Class | DMR | Sham | Overall |
|---|---|---|---|
| Preferred Term | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 Recorded Diabetic History | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Type 2 Diabetes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Prior Therapy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Diabetic Retinopathy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Diabetic Nephropathy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Diabetic Neuropathy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; PT = Preferred Term; SOC = System Organ Class. Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Diabetic histories were coded using MedDRA version 22.0. Subjects were counted once for each system organ class (SOC) and once for each preferred term (PT). Diabetic history terms are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. SOURCE: Listing 16.2.4.2.1





Table 14.1.3.3 Summary of Targeted Hypoglycemic Events History by Treatment Safety Population

| Hypoglycemic Event Number of Events in Past Year Statistic | DMR<br>(N=XX) | Sham<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| real statistic | (14-703) | (14-704) | (14-704) |
| Subjects with at least 1 hypoglycemic event in the past year | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Loss of consciousness | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Admission to hospital | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Seizure | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | xx.x | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1. SOURCE: Listing 16.2.4.2.3

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.1.4 Summary of Prior Medications by ATC Class Level 4, PT, and Treatment Safety Population

| ATC Class Level 4 | DMR | Sham | Overall |
|---|---|---|---|
| Preferred Term (ATC Class Level 5) | (N=XX) | (N=XX) | (N=XX) |
| Subjects with at least 1 Prior Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Prior Diabetic Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Prior Rescue Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Prior Non-Drug Therapy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | | | |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | | | |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ATC = Anatomical Therapeutic Chemical; DMR = duodenal mucosal resurfacing; PT = Preferred Term; WHO-DD = World Health Organization drug dictionary. Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. All medications (concomitant medications, diabetic medications, rescue medications, and non-drug therapies) were coded using WHO-DD version March 2019. Prior medications are all medications (including diabetic medications, rescue medications, and non-drug therapies) that were started before the index procedure whether or not they were stopped before the index procedure. Medications are displayed by descending frequency of ATC Level 4 classification, by PT within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT. SOURCE: Listing 16.2.8.6

**Programming note:** Ensure proper WHO-DD version is displayed in footnote.





#### Table 14.1.5.1 Summary of Endoscopic Evaluation Medication Run-In Population

Visit: Baseline

| Variable | DMR | Sham | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Grade of Esophagitis | | | |
| None | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Grade 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Grade 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Duodenum Accessed | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Furthest Location Accessed | | | |
| D1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormalities of GI Tract Preventing Access to Duodenum | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Anatomic abnormalities Precluding Completion of DMR | | | |
| Procedure | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; GI = gastrointestinal.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

SOURCE: Listing 16.2.5.3.3

Programming note: Repeat for Week 24 for cross-over subjects. Only Sham and Overall columns will be included at this visit.





# Table 14.1.5.1 (cont.) Summary of Endoscopic Evaluation Medication Run-In Population

Visit: Baseline

| Variable | DMR | Sham | Overall |
|---------------------------------------|------------|------------|------------|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| GI Conditions | | | |
| Bleeding | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ulcer(s) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Varices() | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Stricture(s) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Telangiectasia | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Malignancy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Endoscopy Successfully Completed | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Excluded Based on Endoscopic Findings | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; GI = gastrointestinal.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

SOURCE: Listing 16.2.5..3.3

Programming note: Repeat for Week 24 for cross-over subjects. Only Sham and Overall columns will be included at this visit.





#### Table 14.1.5.2 Summary of Endoscopy Results Safety Population

Visit: Baseline

| Variable<br>Statistic or Category | DMR<br>(N=XX) | Sham<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Statistic of Gategory | (N-XX) | (14-///) | (14-XX) |
| Ulcers Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Luminal Narrowing Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| D4 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Length of Luminal Narrowing | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Diameter of Luminal Narrowing | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 - Q1. SOURCE: Listing 16.2.5.3.4





# Table 14.1.5.2 (cont.) Summary of Endoscopy Results Safety Population

| ١ | /isi | t: E | 3as | elir | ıе |
|---|------|------|-----|------|----|

| Variable | DMR | Sham | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Visual Appearance D1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Partial Regrowth | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reduction in Height and/or Width of Plicae | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Bleeding Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other Mucosal Abnormality | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Visual Appearance D2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Partial Regrowth | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reduction in Height and/or Width of Plicae | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Bleeding Present | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other Mucosal Abnormality | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Continue for D3 and D4 Findings

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1.

SOURCE: Listing 16.2.5.3.4

Programming note: Repeat for Week 24 for cross-over subjects. Only Sham and Overall columns will be included at this visit.





#### Table 14.2.1.1 Summary of Change from Baseline in HbA1c by Study Visit and Treatment AT Population

| Study Visit | DMR<br>(N=XX) | | Sham<br>(N=XX) | | | |
|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | %CFB | Observed | CFB | %CFB |
| Baseline [1] | | | | | | |
| n | XX | | | XX | | |
| Mean (SD) | XX.X (XX.XX) | | | XX.X (XX.XX) | | |
| 95% CI of the Mean | (XX.X, XX.X) | | | (XX.X, XX.X) | | |
| Median | XX.X | | | XX.X | | |
| Q1, Q3 | XX, XX | | | XX, XX | | |
| IQR | XX.X | | | XX.X | | |
| Min, Max | XX, XX | | | XX, XX | | |
| | | Repea | t for Week 4, Week 12, and | Week 18. | | |
| Week 24 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| 95% CI of the Mean | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| IQR | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Repeat for Week 36 and Week 48 for DMR only. Repeat for Crossover Week 4, Crossover Week 12, Crossover Week 18, and Crossover Week 24 for Sham only.

Abbreviations: AT = as treated; CFB = change from baseline; IQR = interquartile range.

Note: Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1.

[1] Baseline is defined as the last observation recorded prior to the attempted treatment with index procedure.

SOURCE: Listing 16.2.6.1

Programming note: Check normality per Section 8 of the SAP. If the data are non-normal, use the Wilcoxon signed-rank test and update the footnote accordingly.





#### Table 14.2.1.2 Summary of Change from Baseline in HbA1c by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

Programming note: Add ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment."

Table 14.2.1.3
Summary of Change from Baseline in HbA1c by Study Visit and Treatment
Weel 24 Per Protocol Population

Same shell as 14.2.1.1

Table 14.2.1.4
Summary of HbA1c During Medication Run-In
Medication Run-In Population

#### Same shell as 14.2.1.1

**Programming note:** Remove AT from abbreviations. Update Note: to read "Subjects are summarized overall." Only one treatment group column, Overall, will be displayed. Only Screening and Baseline visits will be displayed and only the observed values will be displayed, no CFB or %CFB columns.





# Table 14.2.1.5 Summary of Change from Week 24 in HbA1c by Study Visit and Treatment AT Population

| Study Visit | Sham<br>(N=XX) | | |
|--------------------|----------------|--------------|--------------|
| Statistic | Observed | Change [1] | % Change [1] |
| Week 24 [2] | | | |
| n | XX | | |
| Mean (SD) | XX.X (XX.XX) | | |
| 95% CI of the Mean | (XX.X, XX.X) | | |
| Median | `XX.X | | |
| Q1, Q3 | XX, XX | | |
| IQR | XX.X | | |
| Min, Max | xx, xx | | |
| Crossover Week 4 | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| 95% CI of the Mean | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

#### Repeat for Crossover Week 12, Crossover Week 18, and Crossover Week 24.

Abbreviations: AT = as treated; IQR = interquartile range.

Note: Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Only Sham cross-over subjects are presented. IQR = Q3 – Q1.

[1] Change from Week 24

[2] The Week 24 value is the value recorded prior to the attempted treatment with the cross-over procedure.

SOURCE: Listing 16.2.6.1

**Programming note:** Check normality per Section 8 of the SAP. If the data are non-normal, use the Wilcoxon signed-rank test and update the footnote accordingly.





#### Table 14.2.1.6 Summary of Change from Week 24 in HbA1c by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.5

Programming note: Add ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Only sham cross-over subjects are presented."





Table 14.2.1.7
Summary of HbA1c Improvement by Study Visit and Treatment
AT Population

| Study Visit | DMR | Sham |
|---------------------|------------|------------|
| Statistic [1] | (N=XX) | (N=XX) |
| Baseline to Week 4 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | xx (xx.x%) |
| Baseline to Week 8 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | XX (XX.X%) |
| Baseline to Week 12 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | XX (XX.X%) |
| Baseline to Week 24 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | xx (xx.x%) |
| Baseline to Week 36 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | xx (xx.x%) |
| Baseline to Week 48 | | |
| Improvement | XX (XX.X%) | XX (XX.X%) |
| No Improvement | XX (XX.X%) | XX (XX.X%) |
| Week 24 to Week 48 | | |
| Improvement | XX (XX.X%) | |
| No Improvement | XX (XX.X%) | |

Abbreviations: AT = as treated.

Note: Subjects are summarized by initial treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. An improvement in HbA1c is defined as any value lower than baseline. The proportion of subjects with an HbA1c improvement at Week 48 is presented for DMR subjects only.

SOURCE: Listing 16.2.6.1





# Table 14.2.1.8 Summary of HbA1c Improvement by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.7

Programming note: Add ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment."

Table 14.2.1.9
Summary of HbA1c Improvement by Study Visit and Treatment
Week 24 PP Population

Same shell as 14.2.1.7





# Table 14.2.2.1 Summary of Change from Baseline in FPG by Study Visit and Treatment AT Population

#### Same shell as 14.2.1.1

Programming note: Add FPG (fasting plasma glucose) to abbreviations. Update SOURCE to Listing 16.2.6.2

Table 14.2.2.2 Summary of Change from Baseline in FPG by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

Programming note: Add FPG (fasting plasma glucose) and ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Update SOURCE to Listing 16.2.6.2




Table 14.2.2.3
Summary of Change from Week 24 in FPG by Study Visit and Treatment AT Population

### Same shell as 14.2.1.5

Programming note: Add FPG (fasting plasma glucose) to abbreviations. Update SOURCE to Listing 16.2.6.2

Table 14.2.2.4 Summary of Change from Week 24 in FPG by Study Visit and Treatment ITT Population

### Same shell as 14.2.1.5

Programming note: Add FPG (fasting plasma glucose) and ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Only Sham cross-over subjects are presented." Update SOURCE to Listing 16.2.6.2





## Table 14.2.3.1 Summary of Change from Baseline in UACR by Study Visit and Treatment AT Population

### Same shell as 14.2.1.1

Programming note: Add UACR (Urine Albumin-to-Creatinine Ratio) to abbreviations. Update SOURCE to Listing 16.2.6.3

Table 14.2.3.2 Summary of Change from Baseline in UACR by Study Visit and Treatment ITT Population

## Same shell as 14.2.1.1

**Programming note:** Add UACR (Urine Albumin-to-Creatinine Ratio) and ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Update SOURCE to Listing 16.2.6.3





## Table 14.2.4.1 Summary of Change from Baseline in ALT by Study Visit and Treatment AT Population

#### Same shell as 14.2.1.1

Programming note: Add ALT (Alanine Aminotransferase) to abbreviations. Update SOURCE to Listing 16.2.6.4

Table 14.2.4.2 Summary of Change from Baseline in ALT by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

**Programming note:** Add ALT (Alanine Aminotransferase) and ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment." Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment."

Update SOURCE to Listing 16.2.6.4





## Table 14.2.5.1 Summary of Change from Baseline in AST by Study Visit and Treatment AT Population

## Same shell as 14.2.1.1

Programming note: Add AST (Aspartate Aminotransferase) to abbreviations. Update SOURCE to Listing 16.2.6.5

Table 14.2.5.2 Summary of Change from Baseline in AST by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

**Programming note:** Add AST (Aspartate Aminotransferase) and ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment."

Update SOURCE to Listing 16.2.6.5





Table 14.2.6.1
Summary of Change from Baseline in SF-36 Scale Scores by Study Visit and Treatment AT Population

### Same shell as 14.2.1.1

Programming note: Update footnote [1] to replace HbA1c with scale score. Include a row at the top of the table "Scale Score: XXXXX". Scale scores will be: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Study visits will include Baseline, Week 12, Week 24, and Week 48 for DMR and Baseline Week 12, Week 24, Crossover week 12 and Crossover Week 24 for Sham. Update SOURCE to Listing 16.2.6.6

Table 14.2.6.2
Summary of Change from Baseline in SF-36 Scale Scores by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

Programming note: Add ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Update footnote [1] to replace HbA1c with scale score. Include a row at the top of the table "Scale Score: XXXXX". Scale scores will be: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Study visits will include Baseline, Week 12, Week 24, and Week 48 for DMR and Baseline Week 12, Week 24, Crossover week 12 and Crossover Week 24 for Sham. Update SOURCE to Listing 16.2.6.6





## Table 14.2.7.1 Summary of Change from Baseline in PROMIS Scores by Study Visit and Treatment AT Population

### Same shell as 14.2.1.1

Programming note: Update footnote [1] to replace HbA1c with score. Include a row at the top of the table "Parameter: XXXXX". Parameters will be: Gastrointestinal Nausea and Vomiting Total Score, Gastrointestinal Gas and Bloating Total Score, Gastrointestinal Diarrhea Total Score, and Belly Pain Total Score. Study visits will include Baseline, Week 12, Week 24, and Week 48 for DMR and Baseline Week 12, Week 24. Crossover week 12 and Crossover Week 24 for Sham. Update SOURCE to Listing 16.2.6.7

Table 14.2.7.2
Summary of Change from Baseline in PROMIS Scores by Study Visit and Treatment ITT Population

#### Same shell as 14.2.1.1

Programming note: Add ITT (Intent-to-Treat) to abbreviations. Update Note: to read "Subjects are summarized by randomized treatment. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment." Update footnote [1] to replace HbA1c with score. Include a row at the top of the table "Parameter: XXXXX". Parameters will be: Gastrointestinal Nausea and Vomiting Total Score, Gastrointestinal Gas and Bloating Total Score, Gastrointestinal Diarrhea Total Score, and Belly Pain Total Score. Study visits will include Baseline, Week 12, Week 24, and Week 48 for DMR and Baseline Week 12, Week 24, Crossover week 12 and Crossover Week 24 for Sham. Update SOURCE to Listing 16.2.6.7





## Table 14.3.1.1 Summary of Adverse Events by Treatment Safety Population

Period: Day 1 - Week 24

| Category | DMR<br>(N=XX) | Sham<br>(N=XX) | Crossover DMR [2]<br>(N=XX) | Combined DMR [3]<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an SAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Maximum Severity of TEAE Mild Moderate Severe | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| Subjects with a TEAE Related to Study Procedure [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE Related to Study Device [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE Leading to Discontinuation of Study | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a TEAE leading to Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a SAE Related to Study Procedure [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with a SAE Related to Study Device [1] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with an UADE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| subjects with an AESI | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: AESI = adverse event of special interest; CI = confidence interval; CRF = case report form; DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event; SAE = serious adverse event; UADE = unanticipated adverse device effect.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and by crossover treatment received. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. AEs were coded using MedDRA version 22.0. A TEAE is any AE with an onset date/time or worsening after DMR or sham procedure.

- [1] Related TEAEs are those marked as Possibly Related, Probably Related, or Definitely Related on the CRF.
- [2] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Day 1 to Week 24 is based on the second procedure.
- [3] Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure. SOURCE: Listing 16.2.7.1

**Programming note:** Repeat for Period: Week 24 – Week 48 where only DMR treatment group column will be displayed and repeat for Day 1 – Week 48 where only Overall treatment group column will be displayed. Ensure proper MedDRA version is printed in the footnote.





Table 14.3.1.2
Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment Safety Population

| | | Day 1 | - Week 24 | | Week 24 - Week 48 | Day 1 - Week 48 |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | DMR<br>(N=XX) | Sham<br>(N=XX) | Crossover DMR [1]<br>(N=XX) | Combined DMR [2]<br>(N=XX) | DMR<br>(N=XX) | Overall (N=XX) |
| Subjects with at least 1<br>TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by crossover treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. AEs were coded using MedDRA version 22.0. A TEAE is any AE with an onset date/time or worsening after DMR or sham procedure. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. If a subject has separate AEs with the same SOC/PT with one starting in the double-blind period and the other starting after Week 24, they are counted once within each period.

[1] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Day 1 to Week 24 is based on the second procedure.

SOURCE: Listing 16.2.7.1

Programming note: SOC & PT text should be in proper case. Ensure correct MedDRA version is printed in footnote. If columns are too wide, repeat table by period.



Table 14.3.1.3
Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment Safety Population

| | | Day 1 | - Week 24 | | Week 24 - Week 48 | Day 1 - Week 48 |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term<br>Maximum Severity | DMR Sham (N=XX) | | Crossover DMR [1] Combined DMR [2] (N=XX) (N=XX) | | DMR<br>(N=XX) | Overall<br>(N=XX) |
| Subjects with at least 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | | |
| TEAE | 707 (707.7770) | 70x (70x.7c70) | 70X (70X.77%) | 701 (701.7770) | XX (XX.X%) | XX (XX.X%) |
| Any Event (Total) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | | | | | | |
| Any Event (Total) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Mild | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Moderate | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Severe | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. AEs were coded using MedDRA version 22.0. A TEAE is any AE with an onset date/time or worsening after DMR or sham procedure. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. If a subject has separate AEs with the same SOC/PT with one starting in the double-blind period and the other starting after Week 24, they are counted once within each period.

Programming note: SOC & PT text should be in proper case. Ensure correct MedDRA version is printed in footnote. If columns are too wide, repeat table by period.

<sup>[1]</sup> Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Day 1 to Week 24 is based on the second procedure.

<sup>[2]</sup> Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure. SOURCE: Listing 16.2.7.1



Table 14.3.1.4 Incidence of Treatment Emergent Adverse Events by Relationship, SOC, PT, and Treatment Safety Population

| | | Day | 1 - Week 24 | | Week 24 - Week 48 | Day 1 - Week 48 |
|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term<br>Maximum Severity | DMR<br>(N=XX) | Sham<br>(N=XX) | Crossover DMR [1]<br>(N=XX) | Combined DMR [2]<br>(N=XX) | DMR<br>(N=XX) | Overall<br>(N=XX) |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Any Event (Total) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| System Organ Class 1 | | | | | | |
| Any Event (Total) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Duefermed Terre 4 | VV (VV V0/ ) | VV (VV V0/ ) | VV (VV V0/ ) | VV (VV V0/ ) | VV (VV V0/) | VV (VV V0() |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Device | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Not Related to Procedure | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: CRF = case report form; DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event. Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. AEs were coded using MedDRA version 22.0. A TEAE is any AE with an onset date/time or worsening after DMR or sham procedure. Related TEAEs are those marked as Possibly Related, Probably Related, or Definitely Related on the CRF. Subjects are counted once for each system organ class (SOC) and once for each preferred term (PT). AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. If a subject has separate AEs with the same SOC/PT with one starting in the double-blind period and the other starting after Week 24, they are counted once within each period.

AD-ST-33.05 Effective date: 22-Jan-2018

<sup>[1]</sup> Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Day 1 to Week 24 is based on the second procedure.

<sup>[2]</sup> Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure. SOURCE: Listing 16.2.7.1





Programming note: SOC & PT text should be in proper case. Ensure correct MedDRA version is printed in footnote. If columns are too wide, repeat table by period.

Table 14.3.2.1 Incidence of Adverse Events Leading to Withdrawal by SOC, PT, and Treatment Safety Population

## Same shell as 14.3.1.2

Programming note: Change first row to read "Subjects with at least 1 TEAE Leading to Withdrawal"

Table 14.3.2.2
Incidence of Adverse Events Leading to Withdrawal by Relationship, SOC, PT, and Treatment Safety Population

Same shell as 14.3.1.4

Programming note: Change first row to read "Subjects with at least 1 TEAE Leading to Withdrawal"





## Table 14.3.2.3 Incidence of Serious Adverse Events by SOC, PT, and Treatment Safety Population

## Same shell as 14.3.1.2

Programming note: Change first row to read "Subjects with at least 1 SAE" Add SAE (serious adverse event) to abbreviations.

Table 14.3.2.4
Incidence of Serious Adverse Events by Relationship, SOC, PT, and Treatment Safety Population

## Same shell as 14.3.1.4

Programming note: Change first row to read "Subjects with at least 1 SAE" Add SAE (serious adverse event) to abbreviations.





# Table 14.3.2.5 Incidence of Unanticipated Adverse Device Effects by SOC, PT, and Treatment Safety Population

### Same shell as 14.3.1.2

Programming note: Change first row to read "Subjects with at least 1 UADE" Add UADE (unanticipated adverse device effect) to abbreviations.

Table 14.3.2.6
Incidence of Unanticipated Adverse Device Effects by Relationship, SOC, PT, and Treatment Safety Population

#### Same shell as 14.3.1.4

Programming note: Change first row to read "Subjects with at least 1 UADE" Add UADE (unanticipated adverse device effect) to abbreviations.

Table 14.3.2.7
Incidence of Adverse Events of Special Interest by SOC, PT, and Treatment Safety Population

### Same shell as 14.3.1.2

Programming note: Change first row to read "Subjects with at least 1 AESI" Add AESI (adverse event of special interest) to abbreviations.

Table 14.3.2.8
Incidence of COVID-19 Adverse Events by SOC, PT, and Treatment
Safety Population

#### Same shell as 14.3.1.2

**Programming note:** Change first row to read "Subjects with at least 1 COVID-19 Related AE" Add COVID-19 (coronavirus 2019) to abbreviations. A footnote will be added after AE review occure prior to lock to define the MedDRA preferred terms included in this summary.





Table 14.3.2.9 Summary of Hypoglycemic Events by Treatment Safety Population

| Variable<br>Statistic or Category | DMR<br>(N=XX) | Sham<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|
| Clations of Gategory | (11 700) | (11 700) | (11 701) |
| Reporting Type | | | |
| Patient | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Physician | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) |
| Blood Glucose Value | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Fasting | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Resolved | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Ongoing | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Duration of Episode | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| IQR | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range; SAE = serious adverse event.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1. SOURCE: Listing 16.2.7.2

AD-ST-33.05 Effective date: 22-Jan-2018





## Table 14.3.2.9 (cont.) Summary of Hypoglycemic Events by Treatment Safety Population

| Variable | DMR | Sham | Overall |
|---|---|---|---|
| Statistic or Category | (N=XX) | (N=XX) | (N=XX) |
| Freated | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Freated with | | | |
| Snack or Meal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Glucose Tablets | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Glucagon | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| IV Glucose | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Medical Attention | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Other | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Symptoms | | | |
| Glucose Alert Value (≤70 mg/dL) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Serious, Clinically Important Hypoclycemia (<54 mg/dL) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Hypoglycemia requiring third-party assistance | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Meet Crtieria for SAE | | | |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing; IQR = interquartile range; SAE = serious adverse event.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1. SOURCE: Listing 16.2.7.2





## Table 14.3.2.10 Summary of Diarrhea by Treatment Safety Population

Period: Day 1 - Week 24

| Study Visit | DMR<br>(N=XX) | | Sham<br>(N=XX) | | Crossover DMR [1]<br>(N=XX) | | Combined DMR [2]<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|
| Category | Freq | n (%) | Freq | n (%) | Freq | n (%) | Freq | n (%) |
| Subjects with at least 1 Diarrhea AESI | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |
| Diarrhea Characteristics | | | | | | | | |
| Bloody | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |
| Steatorrhea | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |
| Other Clinical Symptoms | | | | | | | | |
| Fever | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |
| Abdominal Pain | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |
| Other | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) | XX | XX (XX.X%) |

Abbreviation: AESI = adverse event of special interest; DMR = duodenal mucosal resurfacing.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. Freq represents the number of events and n and % represents the number of subjects.

I11 Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure): Baseline to Week 24 is based on the second procedure.

SOURCE: Listing 16.2.7.1

Programming note: Repeat for Period: Week 24 – Week 48 where only DMR treatment group column will be displayed and repeat for Day 1 – Week 48 where only Overall treatment group column will be displayed.

<sup>[2]</sup> Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.





## Table 14.3.3.1 Listing of Adverse Events Leading to Withdrawal All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time (Study Day) | Severity/<br>Relationship to<br>Procedure/<br>Relationship<br>to Device | Device/ | Serious? | TEAE? | UADE? /<br>Medical<br>History<br>Relevant to<br>SAE/UADE | Caused Subject<br>to be<br>discontinued<br>from the study? |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>DDMMMYYYY/HH:MM (X) | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXXX/<br>XXXX | xx | XX | XX/<br>XXX | XX |
| XXXXX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>Ongoing | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXX | Yes: XXXXXX | XXX | XX/<br>XXX | XXX |
| | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>DDMMMYYYY/HH:MM (X) | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXX | XX | XX | XX/<br>XXX | XX |

Abbreviations: DMR = duodenal mucosal resurfacing; GI = gastrointestinal; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event; UADE = unanticipated adverse device effect.

Note: Study day is calculated relative to the date of index procedure. Adverse events were coded using MedDRA version 22.0. A TEAE is any AE that starts or worsens after the start of DMR or Sham procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If time missing, display "- -:- -". If Other Action Taken? is Other or Concomitant Medication, concatenate all specify fields with a semicolon. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." Ensure correct MedDRA version is printed in footnote.





## Table 14.3.3.1 (cont.) Listing of Adverse Events Leading to Withdrawal All Subjects

| Subject<br>ID | | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time (Study<br>Day) | AESI? | Time from<br>DMR/Sham<br>Procedure<br>(Days, Hours | (Days, | If Diarrhea,<br>Characteristics/Other<br>Clinical Symptoms | If GI Bleeding,<br>Add'l Lab or<br>Diagnostic Tests<br>Conducted? | Cause for<br>Fever/Add'l<br>Symptoms | Other<br>Additional<br>Symptoms |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx | XXXXXXXXXXXXX | DDMMMYYYY/HH:MM<br>(X) /<br>DDMMMYYYY/HH:MM<br>(X) | | XX, XX | XX, XX | XXXXX/XXXXX | XX | XXXXX/XXXXX | XXXXX |
| XXXXX | xxxxx | XXXXXXXXXXXXX | DDMMMYYYY/HH:MM<br>(X)<br>/Ongoing | XXX;XXXXXX | XXX, XX | XX, XX | XXXXX | XXX | xxxxx | xxxxx |
| | XXXXX | | DDMMMYYYY/HH:MM | | XX, XX | XX, XX | XXXXX/XXXXX | XX | XXXXX/XXXX | XXXXX |

Abbreviation: AESI = adverse event of special interest; DMR = duodenal mucosal resurfacing; GI = gastrointestinal; TEAE = treatment emergent adverse event; UADE = unanticipated adverse device effect.

Note: Study day is calculated relative to the date of index procedure. Adverse events were coded using MedDRA version 22.0. A TEAE is any AE that starts or worsens after the start of DMR or Sham procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

Programming note: Ensure proper MedDRA version is displayed in footnote.





Table 14.3.3.2 Listing of Serious Adverse Events Safety Population

Same shell as 14.3.3.1

Table 14.3.3.3 Listing of Deaths Safety Population

Same shell as 14.3.3.1

Table 14.3.3.4 Listing of Unanticipated Adverse Device Effects Safety Population

Same shell as 14.3.3.1

Table 14.3.3.5 Listing of Adverse Events of Special Interest Safety Population

Same shell as 14.3.3.1





## Table 14.3.4.1 Listing of Abnormal Laboratory Data Safety Population

| Subject<br>ID | Randomized<br>Treatment [1] | Parameter (unit) | Study<br>Visit | Date of<br>Collection<br>(Study Day) | Standard<br>Results | Change<br>from<br>Baseline<br>[3] | Reference<br>Range<br>[4] | Reference<br>Range Flag | Accession<br>Number | Abnormally<br>Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXX | Hematocrit (unit) | xxxxxx | DDMMMYYYY<br>(X) | XX | | XX – YY | | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | XXX | XXXXXX | XX |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXX | |
| | | | XXXXXX | (X) | ND | | | | | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXXX | |

Abbreviations: A = abnormal; DMR = duodenal mucosal resurfacing; H = high; L = low.

Note: Study day is calculated relative to the date of index procedure.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

<sup>[2]</sup> Baseline is the last measurement taken before the index procedure.

<sup>[3]</sup> Reference range is used to identify potentially clinically significant laboratory values.





Table 14.3.5.1.1
Summary of Complete Blood Count Laboratory Results by Study Visit and Treatment
Safety Population

Period: Baseline - Week 24

| Parameter (unit)<br>Study Visit | DMR<br>(N=XX) | | Sham<br>(N=XX) | | Crossover DMR [2]<br>(N=XX) | | Combined DMR [3]<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | Observed | CFB | Observed | CFB | Observed | CFB |
| Hematocrit (unit) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| n | XX | | XX | | XX | | XX | |
| Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| Median | XX.X | | XX.X | | XX.X | | XX.X | |
| Q1, Q3 | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| IQR | XX.X | | XX.X | | XX.X | | XX.X | |
| Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| Week 4 | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | | XX.X | | XX.X | | XX.X | | XX.X |
| | XX.X (XX.XX) | (XX.XX) | XX.X (XX.XX) | (XX.XX) | XX.X (XX.XX) | (XX.XX) | XX.X (XX.XX) | (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| IQR | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Abbreviation: CFB = change from baseline; DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1.

- [1] Baseline is defined as the last observation recorded prior to the attempted treatment with index procedure.
- [2] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Baseline to Week 24 is based on the second procedure.
- [3] Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.
- [4] For subjects with index Sham procedure; relative to crossover DMR procedure, which occurred within 21 days from Week 24.

SOURCE: Listing 16.2.8.1.1

Programming Note: Continue for Visits: Week 12, Week 18, Week 24, Week 36, Week 48 and all other parameters. Repeat for period: Week 24 - Week 48 where only the DMR treatment group column will be displayed and for Period: Baseline – Week 48, where only Overall treatment group column will be displayed. For the Baseline – Week 48 table, first column of shell will be further divided by idex/crossover procedure. Shell will be as follows:





## Table 14.3.5.1.1 (cont.) Summary of Complete Blood Count Laboratory Results by Study Visit and Treatment Safety Population

| Oulcity I to | Spaidtion | |
|----------------------------|-----------------|---------|
| Period: Baseline – Week 48 | | |
| Parameter (unit) | Overal | |
| Study Visit | (N=XX | |
| Statistic | Observed | CFB |
| Hematocrit (unit) | | |
| Index DMR or Sham | | |
| Baseline [1] | | |
| n n | XX | |
| Mean (SD) | XX.X (XX.XX) | |
| | XX.X | |
| Week 24 | | |
| n | XX | XX |
| Mean (SD) | VOV.V. (AAV.VA) | XX.X |
| | XX.X (XX.XX) | (XX.XX) |
| Index DMR | | |
| Week 36 | | |
| n | XX | XX |
| Mean (SD) | ,,,, | XX.X |
| | XX.X (XX.XX) | (XX.XX) |
| ••• | · · · · | , |
| Week 48 | | |
| n<br>Maria (OD) | XX | XX |
| Mean (SD) | VV V (VV VV) | XX.X |
| | XX.X (XX.XX) | (XX.XX) |
| Crossover DMR [4] | | |
| Crossover Week 4 | | |
| n | XX | XX |

Abbreviation: CFB = change from baseline; DMR = duodenal mucosal resurfacing; IQR = interquartile range.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. IQR = Q3 – Q1.

- [1] Baseline is defined as the last observation recorded prior to the attempted treatment with index procedure.
- [2] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Baseline to Week 24 is based on the second procedure.
- [3] Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.
- [4] For subjects with index Sham procedure; relative to crossover DMR procedure, which occurred within 21 days from Week 24.

SOURCE: Listing 16.2.8.1.1

AD-ST-33.05 Effective date: 22-Jan-2018





Table 14.3.5.1.2
Shift from Baseline in Complete Blood Count Laboratory Results by Study Visit and Treatment Safety Population

Period: Baseline - Week 24

| | | Baselin | e [1] | |
|---|---|---|---|---|
| Parameter | | DMR (N | =XX) | |
| Study Visit<br>Category | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) |
| Hematocrit (unit) | | | | |
| Week 4 | | | | |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 12 | | | | |
| Low | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| High | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: DMR = duodenal mucosal resurfacing.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

- [1] Baseline is defined as the last observation recorded prior to the attempted treatment with index procedure
- [2] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Baseline to Week 24 is based on the second procedure.
- [3] Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.

SOURCE: Listing 16.2.8.1.1

**Programming Note:** Continue for Visits: Week 18, Week 24, Week 36, Week 48 and all other parameters. Repeat for DMR, Sham, Crossover DMR [2], and Combined DMR [3] treatment groups for period: Baseline – Week 24. Repeat for period: Week 24 - Week 48 where only the DMR treatment group column will be displayed and for Period: Baseline – Week 48, where only Overall treatment group column will be displayed and the first column will be further divived by index/crossover procedure. Sort alphabetically by parameter.





Table 14.3.5.2.1 Summary of Blood Chemistry Laboratory Results by Study Visit and Treatment Safety Population

### Same shell as 14.3.5.1.1

Programming note: Update SOURCE to Listing 16.2.8.1.2.

Table 14.3.5.2.2
Shift from Baseline in Blood Chemistry Laboratory Results by Study Visit and Treatment Safety Population

### Same shell as 14.3.5.1.2

Programming note: Update SOURCE to Listing 16.2.8.1.2.

Table 14.3.5.3.1 Summary of Urinalysis Laboratory Results by Study Visit and Treatment Safety Population

## Same shell as 14.3.5.1.1

Programming note: Update SOURCE to Listing 16.2.8.1.3.

Table 14.3.5.3.2
Shift from Baseline in Urinalysis Laboratory Results by Study Visit and Treatment Safety Population

#### Same shell as 14.3.5.1.2

Programming note: Update SOURCE to Listing 16.2.8.1.3.





## Table 14.3.6.1.1 Summary of Vital Signs by Study Visit and Treatment Safety Population

### Same shell as 14.3.5.1.1

Programming note: Visits include Screening, Baseline, Week 4, Week 12, Week 18, Week 24, Week 36, and Week 48. Parameters include weight (kg), sitting systolic blood pressure (mmHg), and pulse rate (bpm). Update SOURCE: to Listing 16.2.8.2

Table 14.3.6.2.1 Summary of 12-Lead Electrocardiogram Results by Study Visit and Treatment Safety Population

## Same shell as 14.3.5.1.1

Programming note: Visits include Screening and Week 24. Parameters include PR interval (msec), RR interval (msec), ventricular rate (bpm), QRS interval (msec), uncorrected QT interval (ms), and QTcB interval (ms). Update SOURCE: to Listing 16.2.8.3





Table 14.3.6.2.2 Summary of 12-Lead Electrocardiogram Interpretation by Study Visit and Treatment Safety Population

| | | Baselir | ne - Week 24 | | Week 24 - Week 48 | Baseline - Week 48 |
|---|---|---|---|---|---|---|
| Study Visit<br>Category | DMR<br>(N=XX) | Sham<br>(N=XX) | Crossover DMR [2]<br>(N=XX) | Combined DMR [3]<br>(N=XX) | DMR<br>(N=XX) | Overall (N=XX) |
| Corponing | | | | | | |
| Screening<br>Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | VV (VV V0/ ) | VV (VV V0/) |
| | , | ` , | ` , | ' | XX (XX.X%) | XX (XX.X%) |
| Abnormal, NCS | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal, CS | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Week 24 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Normal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal, NCS | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Abnormal, CS | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: CS = clinically significant; DMR = duodenal mucosal resurfacing; NCS = not clinically significant.

Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, by cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR

SOURCE: Listing 16.2.8.3

<sup>[1]</sup> Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Baseline to Week 24 is based on the second procedure.

<sup>[2]</sup> Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.





## Table 14.3.6.3.1 Summary of Concomitant Medications by Treatment Safety Population

| | Day 1 - Week 24 | | | |
|---|---|---|---|---|
| ATC Class Level 4 Preferred Term (ATC Class Level 5) | DMR<br>(N=XX) | Sham<br>(N=XX) | Cross-over DMR [1]<br>(N=XX) | Combined DMR [2]<br>(N=XX) |
| Subjects with at least 1 Concomitant Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Diabetic<br>Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Rescue<br>Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Subjects with at least 1 Non-Drug<br>Therapy | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 1 Preferred Term 2 | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ATC Class 2 | | | | |
| Preferred Term 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Abbreviations: ATC = Anatomical Therapeutic Chemical; DMR = duodenal mucosal resurfacing; PT = Preferred Term; WHO-DD = World Health Organization drug dictionary. Note: Percentages are n/Number of subjects in the Safety Population\*100. Subjects are summarized by initial treatment received, cross-over treatment received, and overall. Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. All medications (concomitant medications, diabetic medications, rescue medications, and non-drug therapies) were coded using WHO-DD version March 2019. Concomitant medications are all medications (including diabetic medications, rescue medications, and non-drug therapies) that were continuing or starting after the index procedure. Medications are displayed by descending frequency of ATC Level 4 classification, by PT within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT.

[1] Subjects who initially received the Sham procedure but received the DMR at Week 24 (relative to index procedure); Day 1 to Week 24 is based on the second procedure.

[2] Subjects who initially received the DMR procedure combined with subjects who initially received the Sham procedure but crossed over to receive the DMR procedure.SOURCE: Listing 16.2.8.6

**Programming note:** Repeat for period: Week 24 - Week 48 where only the DMR treatment group column will be displayed and for Period: Baseline – Week 48, where only Overall treatment group column will be displayed.





## 14.3. Planned Listing Shells

Listing 16.2.1 Subject Disposition All Subjects

| Subject ID | Randomized<br>Treatment<br>[1] | Date of<br>Informed<br>Consent<br>(Study Day) | Subject's<br>Status | Date of<br>Discontinuation/<br>Completion<br>(Study Day) | Reason for<br>Early Termination | Blind Broken? | Was the Subject<br>Unblinded? | Crossover and undergo DMR procedure? |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | DDMMMYYYY<br>(XX) | XXXXXX | DDMMMYYYY (XX) | XXXXXX | XX | XXX | XX |
| XXXXXX | XXXXXX | DDMMMYYYY<br>(XX) | xxxxxx | DDMMMYYYY (XX) | Other: XXXXXXXX | XX | XXX | XX |
| XXXXXX | XXXXXX | DDMMMYYYY<br>(XX) | xxxxxx | DDMMMYYYY (XX) | XXXXXX | Yes:<br>DDMMMYYYY,<br>XXXXXX | XXX | XXX |
| xxxxx | xxxxxx | DDMMMYYYY<br>(XX) | xxxxxx | DDMMMYYYY (XX) | Lost to Follow-up:<br>DDMMMMYYYY | XX | XXX | xxx |
| xxxxx | XXXXXX | DDMMMYYYY<br>(XX) | xxxxxx | DDMMMYYYY (XX) | xxxxxx | XX | XX; XXXXX | xx |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

**Programming Note:** If reason for early termination is Other, concatenate the specify text as shown with a semicolon. If reason for early termination is Lost to Follow-up, concatenate date of last contact as shown with a semicolon. If the Blind was broken, concatenate date the blind was broken and reason for breaking the blind as shown with a semicolon. If the subject was not unblinded, concatenate the Why field with a semicolon.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





## Listing 16.2.2.1 Inclusion and Exclusion Criteria Not Met All Subjects

| Subject ID | Randomized<br>Treatment [1] | Date of Informed Consent<br>(Study Day) | Visit | Visit Date<br>(Study Day) | All Inclusion<br>Criteria Met?<br>[2] | Any Exclusion<br>Criteria Met?<br>[3] |
|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | DDMMMYYYY<br>(-X) | Screening | DDMMMYYYY (-X) | | |
| | | DDMMMYYYY<br>(-X) | Baseline | | No: 02 | No |
| xxxxxx xxxxxx | DDMMMYYYY<br>(-X) | Screening | DDMMMYYYY (-X) | No: 02 | No | |
| | | DDMMMYYYY<br>(-X) | Baseline | | Yes | Yes: 02 |
| XXXXXX | XXXXXX | DDMMMYYYY<br>(-X) | Screening | DDMMMYYYY (-X) | Yes | No |
| | | DDMMMYYYY<br>(-X) | Baseline | | Yes | No |

Abbreviations: DMR = duodenal mucosal resurfacing; IE = inclusion/exclusion.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

IE Description:

Inclusion Criteria:

02 = Diagnosed with T2D for at least 3 years.

Exclusion Criteria:

02 = History of diabetic ketoacidosis or hyperosmolar nonketotic coma.

**Programming note:** If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown in the example. If no criteria are present for a column, remove the [2] and/or [3] from the column header.





## Listing 16.2.2.2.1 Protocol Deviations All Subjects

| | Randomize | d | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | E (B) (" ): | Violation | | Event Date | Date | Action/ | • | IRB Submission | |
| ID | [1] | Event Relationship | Level | Description | (Visit) | Identified | Resolution | IRB | Date | Comments |
| xxxxx | xxxxxx | xxxxxxxxxx | MAJOR | XXXXXXX | DDMMMYYY<br>(XXXXX) | DDMMMYYY | XXXXXXX | XX | DDMMMYYY | XXXXX |
| | | XXXXXXXXXXXX | MINOR | XXXXXXXXXXXXX | DDMMMYYY<br>(XXXXX) | DDMMMYYY | XXXXXXX | XX | DDMMMYYY | XXXXX |
| XXXXXX | xxxxxx | XXXXXXXXXX | MINOR | xxxxxxxxxxxxxxxxx | DDMMMYYY<br>(XXXXX) | DDMMMYYY | XXXXXX | XX | DDMMMYYY | xxxxx |
| | | XXXXXXXXXXXXXXXX | MINOR | XXXXXXXXXX | | | | | | |
| XXXXX | xxxxxx | xxxxxxxxxx | MAJOR | xxxxxxxxxxxxxxxxx | X DDMMMYYY<br>(XXXXX) | DDMMMYYY | xxxxxx | xx | DDMMMYYY | xxxxx |

Abbreviation: DMR = duodenal mucosal resurfacing.

Programming note: The structure of this listing may change depending on the information in the protocol deviations file.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects have the opportunity to crossover and receive DMR treatment.





Listing 16.2.2.2.2 COVID-19 Protocol Deviations All Subjects

Same shell as listing 16.2.2.2.1

Programming note: Add COVID-19 (coronavirus 2019) to abbreviatons.





## Listing 16.2.3 Analysis Populations All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Study<br>[2] | Screened<br>[3] | Medication<br>Run-In<br>[4] | ITT<br>[5] | AT<br>[6] | Reason(s) for Exclusion |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | Yes | Yes | Yes | No | No | ITT; Was not randomized |
| XXXXXX | xxxxxx | Yes | Yes | Yes | Yes | Yes | |
| XXXXXX | XXXXXX | No | No | No | No | No | AT; Did not receive the index procedure |

Abbreviations: AT = as treated; ITT = Intent-to-Treat.

Programming note: Concatenate all reasons for exclusion with a semicolon.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects have the opportunity to crossover and receive DMR treatment.

<sup>[2]</sup> The study population includes all subjects consented at the site.

<sup>[3]</sup> The Screened population includes all subjects who completes Visit 1.

<sup>[4]</sup> The Medication Run-In population includes all subjects who entered the Run-In Phase.

<sup>[5]</sup> The ITT population includes all subjects who were randomized after the Medication Run-In phase.

<sup>[6]</sup> The AT population includes a subset of ITT subjects who received at least one ablation or undergo the randomized sham procedure.





## Listing 16.2.4.1 Demographics and Baseline Characteristics All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Date IC<br>Signed<br>(Study Day)/<br>Re-consent<br>Date<br>(Study Day) | IC Version/<br>Protocol<br>Version/Verify<br>taking 2 or 3<br>OADs? | Sex | Child-<br>Bearing<br>Age? | Date of<br>Birth/<br>Age<br>(years) | Ethnicity | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m²) | Instructed<br>to Begin<br>4-Week<br>Run-In? | Nutrition and<br>Exercise<br>Guidance/<br>Glycemia<br>Diary/Glucose<br>Meter |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxxxx | DDMMMYYYY<br>(XX) | XXX/<br>XXXX/<br>XX | XXXX | XX | DDMMMYYY/<br>XX | XXXXXXX | XXXXXXX | XX.X | XX.X | XX.X | XX | XXX/<br>XXX/<br>XXX |
| XXXXXX | xxxxx | DDMMMYYYY<br>(XX)/<br>DDMMMYYYY<br>(XX) | XXX/<br>XXXX/<br>XX | XXXXXX | XX | DDMMMYYY/<br>XX | xxxxxx | XXXXXX | XX.X | XX.X | XX.X | XX | XXX/<br>XXX/<br>XXX |
| XXXXXX | XXXXXX | DDMMMYYYY<br>(XX) | XXX/<br>XXXX/<br>XX | XXXXXX | XX | DDMMMYYY/<br>XX | xxxxxx | XXXXXX | XX.X | XX.X | XX.X | XX | XXX/<br>XXX/<br>XXX |

Abbreviations: BMI = body mass index; DMR = duodenal mucosal resurfacing; IC = informed consent; OAD = oral antidiabetic medication.

Note: Study day is calculated relative to the date of index procedure. Height and weight are the values at Screening.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

Programming Note: If a subject was re-consented, concatenate the date and study day, otherwise leave blank. If subject has multiple races, concatenate them. If a subject was enrolled under protocol version 1 concatenate the answer to "Verified that the Subject is taking two OADs (metformin plus one additional OAD) at least at half maximum labeled dose (or highest tolerated dose) and details have been recorded on the ConMed CRF." in the cell. If a subject was enrolled under protocol version 2, concatenate the answer to "Verified that the Subject is taking two or three OADs (metformin plus two

Additional OAD) at least at half maximum labeled dose (or highest tolerated dose) and details have been recorded on the ConMed CRF." in the cell.





Listing 16.2.4.2.1 Diabetic History All Subjects

| Subject ID | Randomized<br>Treatment [1] | History | System Organ Class/<br>Preferred Term/<br>Verbatim Term | If Prior Therapy,<br>Describe | Onset Date (Study Day)/<br>End Date (Study Day)/ |
|---|---|---|---|---|---|
| XXXXXX | xxxxx | XXXXXX | XXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXX | xxxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| | | xxxxxx | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXX | xxxxxx | MMMYYYY (X)/<br>Ongoing |
| | | xxxxxx | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXX/<br>XXXXXX | xxxxxx | DDMMMYYYY (X)/<br>Ongoing |
| xxxxxx | XXXXXX | xxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities.

Note: Study day is calculated relative to the date of index procedure. Diabetic history was coded using MedDRA version 22.0. Only subjects with diabetic history recorded are listed. [1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





## Listing 16.2.4.2.2 Medical History All Subjects

| Subject ID | Randomized<br>Treatment<br>[1] | System | Status | System Organ Class/<br>Preferred Term/<br>Verbatim Term | If Prior Therapy,<br>Describe | Start Date (Study Day)/<br>End Date (Study Day)/ |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxxxx | XXXXXX | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXXX | xxxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |
| | | XXXXX; XXXXXXXXX | XXXXX; | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | xxxxxx | MMMYYYY (X)/<br>Ongoing |
| | | xxxxxx | xxxxxx | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | xxxxxx | DDMMMYYYY (X)/<br>Ongoing |
| xxxxxx | xxxxxx | xxxxxx | xxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (X) |

Abbreviations: DMR = duodenal mucosal resurfacing; MedDRA = medical dictionary for regulatory activities.

Note: Study day is calculated relative to the date of index procedure. Medical history was coded using MedDRA version 22.0. Only subjects with medical history recorded are listed. [1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** Concatenate 'Specify Other System' field with a semicolon.





## Listing 16.2.4.2.3 Targeted Hypoglycemic Events History All Subjects

| Subject ID | Randomized<br>Treatment<br>[1] | Experienced Hypoglycemic Events in the Past Year? | Event | Check if None | Number of Events in<br>Past Year |
|---|---|---|---|---|---|
| xxxxx | XXXXXX | xxx | Loss of consciousness<br>Admission to hospital<br>Seizure | NONE<br>NONE | X |
| xxxxx | xxxxxx | XXX | Loss of consciousness<br>Admission to hospital<br>Seizure | | X<br>X<br>X |

Abbreviation: DMR = duodenal mucosal resurfacing.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.




#### Listing 16.2.5.1.1 DMR Procedure Pre-Op All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | DMR Procedure<br>Performed? | Administered Paracetamol, Acetaminophen or Equivalent Prior to Procedure? | Procedure Timepoint | Type of<br>Anesthesia/Sedation | Date DMR<br>Procedure<br>Performed<br>(Study Day) | Start Time/End Time |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | XXX | XXXXX | XXXXXXX | DDMMMYYY<br>(XX) | HH:MM/HH:MM |
| XXXXXX | xxxxx | XX; XXXXXX | | | | | |

Abbreviation: DMR = duodenal mucosal resurfacing.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If DMR procedure was not performed, concatenate reason with a semicolon.





# Listing 16.2.5.1.2 DMR Procedure Lift and Ablation Details All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Start Location/<br>End Location | Time Scope In/<br>Time Scope out | Number of<br>Injections/Mucosal<br>Lifts | Number of<br>Ablations | Distance from<br>Papilla to<br>Proximal Edge<br>of First<br>Completed<br>Ablation (cm) | Procedure<br>Successfully<br>Completed? | Fluoroscopy<br>Exposure<br>Duration<br>(minutes) | Radiation due<br>to Fluoroscopy<br>Exposure<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxx | XXXX/XXX | HH:MM / HH:MM | X | X | XXX | XXX | XX | XXX (XXX) |
| xxxxx | xxxxx | XXXX/XXX | HH:MM / HH:MM | X | X | XXX | XX; XXXXX;<br>XXXXXX | xx | XXX (X) |

Abbreviation: DMR = duodenal mucosal resurfacing.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If the procedure was not successfully completed, concatenate the 'No, why?' field in the cell with a semicolon. If the reason was other, also concatenate the 'Specify' field and 'Detail' with a semicolon. Concatenate the Radiation due to Fluoroscopy exposure unit in the cell in parenthesis.





#### Listing 16.2.5.2.1 Sham Procedure Pre-Op All Subjects

| Subject ID | Randomized<br>Treatment [1] | Sham Procedure Performed? | Administered Paracetamol,<br>Acetaminophen or Equivalent<br>Prior to Procedure? | Date DMR Procedure Performed<br>(Study Day) | Type of Anesthesia/Sedation |
|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | XXX | DDMMMYYY<br>(XX) | XXXXXXX |
| xxxxxx | xxxxxx | XX; XXXXXX | | | |

Abbreviation: DMR = duodenal mucosal resurfacing.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If Sham procedure was not performed, concatenate reason with a semicolon.





#### Listing 16.2.5.2.2 Sham Procedure Details All Subjects

| Subject<br>ID<br>XXXXXX | Randomized<br>Treatment<br>[1] | Start Time of Procedure HH:MM | Time of Insertion of Revita Catheter | Time of Removal of<br>the Revita Catheter<br>HH:MM | Total time<br>Catheter<br>Indwelling<br>HH:MM | End Time of<br>Procedure<br>HH:MM | Fluoroscopy<br>Exposure<br>Duration<br>(minutes) | Radiation due to Fluoroscopy Exposure (unit) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | НН:ММ | нн:мм | HH:MM | нн:мм | нн:мм | xx | XXX (XX) |

Abbreviation: DMR = duodenal mucosal resurfacing.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

Programming note: Concatenate the 'Radiation due to Fluoroscopy Exposure Unit' in the cell in parenthesis.





#### Listing 16.2.5.3.1 Device Use Summary All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Type of Procedure | Date of Procedure<br>(Study Day) | Device Type | Not Used | Lot/Serial<br>Number | Device<br>Disposition |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | XXXXX | DDMMMYYY<br>(XX) | Console | | XX-XXXX | XXXXXXXXX |
| | | | · / | Revita Catheter | | XX-XXXX | XXXXXXXXX |
| | | | | Line Set | | XX-XXXX | XXXXXXXXX |
| | | | | HF Umbilical | | XX-XXXX | XXXXXXXXX |
| xxxxx | XXXXXX | XXXXX | DDMMMYYY<br>(XX) | Console | | XX-XXXX | XXXXXXXXX |
| | | | (704) | Revita Catheter | | XX-XXXX | XXXXXXXXXX |
| | | | | Line Set<br>HF Umbilical | Not used | XX-XXXX | XXXXXXXXX |

Abbreviation: DMR = duodenal mucosal resurfacing.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.5.3.2 Device Malfunction All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Any Device<br>Malfunctions | Date of<br>Malfunction<br>(Study Day) | Which<br>Component<br>Malfunctioned? | Lot/Serial<br>Number | At What<br>Point Did<br>the<br>Malfunction<br>Occur? | Describe<br>the Specific<br>Malfunction | Result in AE? | Final Disposition of Malfunctioning Device |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | XXX | DDMMMYYY<br>(XX) | XXXXX | XX-XXXX | XXXXX | XXXXXX | XX | xxxx;xxxx |
| XXXXXX | XXXXXX | XXXXX | DDMMMYYY<br>(XX) | xxxxx | XX-XXXX | XXXXX;<br>XXXXX | XXXXXX | XX | xxxxx |

Abbreviation: DMR = duodenal mucosal resurfacing.

**Programming note:** If the point the malfunction occurred was Other, concatenate the specify field in the cell with a semicolon. If the final disposition is other, concatenate the specify field in the cell with a semicolon.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.5.4.1 Endoscopic Evaluation All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Endoscopic<br>Evaluation<br>Performed? | Date /Time<br>Performed<br>(Study Day) | Presence of<br>Esophagitis/Grade | Duodenum<br>Accessed?/Furthest<br>Location Accessed | Abnormalities<br>Preventing<br>Endoscopic<br>Access? | Abnormalities<br>Precluding<br>Completion<br>of DMR? | Upper GI<br>Conditions? | Endoscopy<br>Successfully<br>Completed? | Excluded<br>Based on<br>Findings? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxxxx | XXX | DDMMMYYY/<br>HH:MM (XX) | XXX / X | XXX / XX | xx | xx | XXX;<br>XXXX,<br>XXXXX | XXX | xx |
| XXXXXX | xxxxxx | XX; XXXXX | DDMMMYYY/<br>HH:MM (XX) | XXX / X | XXX / XX | XXX; XXXX | XXX;XXXX | xx | xx; xxxx | |

Abbreviation: DMR = duodenal mucosal resurfacing.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If the abnormality preventing endoscopic access to the duodenum is Other, concatenate the specify field in the cell with a semicolon. If the abnormality precluding completion of DMR is other, concatenate the specify field in the cell with a semicolon. If GI conditions were identified, concatenate all that apply in the cell separated by a comma. If the GI condition is other, concatenate specify field in cell. If the endoscopy procedure was not successfully completed, concatenate the 'No, explain' field in the cell with a semicolon.

excluded based on endoscopic findings, concatenate the 'Yes, explain' field in the cell with a semicolon.





Listing 16.2.5.4.2 Endoscopy All Subjects

| | | | | | Visual Appearance | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Randomized<br>Treatment<br>[1] | Endoscopy<br>Performed? | Date of<br>Procedure<br>(Study Day) | Location of<br>Endoscopy | Ulcer(s)? /<br>Location | Luminal<br>Narrowing? /<br>Length (mm) /<br>Diameter (mm) | D1 Done? /<br>Findings | D2 Done?<br>/ Findings | D3 Done? /<br>Findings | D4 Done?<br>/ Findings |
| XXXXXX | xxxxxx | xxx | DDMMMYYY<br>(XX) | XX, XX, XX,XX | XXX /<br>XXXX | XXX /<br>XXX /<br>XXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX |
| xxxxxx | xxxxxx | XX; XXXXX | DDMMMYYY<br>(XX) | XX, XX, XX,XX | XXX /<br>XXXX | XXX /<br>XXX /<br>XXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX | XXX /<br>XXXXXX |

Abbreviation: DMR = duodenal mucosal resurfacing.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.5.4.3 Biopsy All Subjects

### Abnormal-Appearing Mucosa

Biopsy Samples Circumferential 4 Quadrant Biopsy Samples Q1 Biopsy Q2 Biopsy Q3 Biopsy Q4 Biopsy Reason Comments Date/Time D1 – Performed Performed Performed Performed Not Randomized Biopsy Biopsy CONTROL from from from from Performed Performed Subject Treatment Sample Successful Biopsy Ablated Ablated Ablated Ablated Endoscopy Performed? (Study Day) Number Location Completion performed Zone? Zone? ID [1] Zone? Zone? XXXXXX XXXXXX XXX DDMMMYYY A1 XX Χ Χ Χ Χ Х Χ XXXXX (XX) A2 XX Χ Х Χ Χ Χ Χ A3 XX Χ Χ Χ Χ Х Χ XXXXXX Х Х Х A4 XX Χ Х Χ XXXXXX XXXXXX XX; XXXXX DDMMMYYY Α1 XX Χ Χ Χ Х Χ Χ (XX) A2 XX Χ Χ Χ Χ Χ Χ А3 XXΧ Χ Χ Χ Χ Χ A4 XX Χ Χ Χ Χ Χ

Abbreviations: DMR = duodenal mucosal resurfacing; Q = quadrant.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.5.5.1 Discharge Information All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Date of<br>Discharge<br>(Study Day) | Procedure<br>Timepoint | Date of First<br>Oral Intake<br>(Study Day) | Any<br>Hypoglycemic<br>events? | Any<br>AEs? | Instructions for 14<br>Day Post-Procedure<br>Diet? | Reminded to Conduct<br>Blood Glucose<br>Monitoring 4x per Day? | Use of OAD<br>Medications<br>Reviewed? |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxxxx | DDMMMYYY<br>(XX) | XXXXX | D DMMMYYY<br>(XX) | XX | XX | XXX | XXX | XXX |

Abbreviations: AE = adverse event; DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.6.1 HbA1c All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | Parameter (unit) | Study<br>Visit | Date of<br>Collection<br>(Study Day) | Standard<br>Results | Change<br>from<br>Baseline<br>[3] | Reference<br>Range<br>[4] | Reference<br>Range Flag | Accession<br>Number | Abnormally<br>Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXX | Hem (unit) | XXXXXX | DDMMMYYYY<br>(X) | XX | | XX – YY | | XXXXXXX | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | XXX | XXXXXX | XX |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXX | |
| | | | XXXXXX | (70) | ND | | | | | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXXX | |

Abbreviations: A = abnormal; DMR = duodenal mucosal resurfacing; H = high; L = low. Note: Study day is calculated relative to the date of index procedure.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

<sup>[2]</sup> Baseline is the last measurement taken before the index procedure.

<sup>[3]</sup> Reference range is used to identify potentially clinically significant laboratory values.





Listing 16.2.6.2
Fasting Plasma Glucose (FPG)
All Subjects

Same shell as 16.2.6.1

Listing 16.2.6.3 Urine Albumin Creatinine Ratio (UACR) All Subjects

Same shell as 16.2.6.1

Listing 16.2.6.4 Alanine Aminotransferase (ALT) All Subjects

Same shell as 16.2.6.1

Listing 16.2.6.5 Aspartate Aminotransferase (AST) All Subjects

Same shell as 16.2.6.1





#### Listing 16.2.6.6 SF-36 Quality of Life Questionnaire All Subjects

| Subject ID | Randomized<br>Treatment [1] | Study Visit | Question | Result |
|---|---|---|---|---|
| xxxxxx | XXXXX | xxxxx | In general, would you say your health is:<br>Compared to one year ago, how would<br>you rate your health in general now?<br>Vigorous Activities, such as running,<br>lifting heavy objects, participating in<br>strenuous sports | XXXXX<br>XXXXX<br>XXXXX |
| | | | Physical functioning scale score Bodily pain scale score scale score Role limitations due to physical health problems scale score Role limitations due to personal or emotional problems scale score Emotional well-being scale score Social functioning scale score Energy/fatigue scale score General health perceptions scale score | XXXXX<br>XXXXX<br>XXXXX<br>XXXXX<br>XXXXX<br>XXXXX<br>XXXX |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Derivations for each of the scale scores are described in Section 6.1.7 of the statistical analysis plan.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





Listing 16.2.6.7 PROMIS Scores All Subjects

| Subject ID | Randomized<br>Treatment [1] | Was Assessment Completed? | Date of Assessment<br>(Study Day) | Question | Result |
|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | XXXXX | How often did you have nausea-that is, a feeling like you could vomit? | XXXXX |
| | | | | How often did you know that you would have nausea before it happened? | XXXXX |
| | | | | How often did you have a poor appetite? | XXXXX |
| | | | | How often did you throw up or vomit? | XXXXX |
| | | | | Gastrointestinal Nausea and Vomiting Total Score | XXXXX |
| | | | | •••• | |

Abbreviations: DMR = duodenal mucosal resurfacing; Patient Reported Outcomes Measurement Information System.

Note: Study day is calculated relative to the date of index procedure.

PROMIS Gastrointestinal Nausea and Vomiting Total Score = sum of the 4 individual items, with a range of 0 to 20, where higher scores indicate worse and more frequent nausea and vomiting.

PROMIS Gastrointestinal Gas and Bloating Total Score = sum of the 13 individual items, with a range of 0 to 65, where higher scores indicate worse and more frequent gas and bloating

PROMIS Gastrointestinal Diarrhea Total Score = sum of the 6 individual items, with a range of 0 to 30, where higher scores indicate worse and more frequent diarrhea. PROMIS Belly Pain Total Score = sum of the 5 individual items, with a range of 0 to 25, where higher scores indicate worse and more frequent belly pain.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

Programming note: If assessment was not completed, concatenate reason in the cell with a semicolon.





Listing 16.2.7.1 Adverse Events All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>(Study Day)/<br>End Date/Time (Study Day) | Severity/<br>Relationship to<br>Procedure/<br>Relationship<br>to Device | Outcome/<br>Action Taken with<br>Device/<br>Other Action<br>Taken | Serious? | TEAE? | UADE? /<br>Medical<br>History<br>Relevant to<br>SAE/UADE | Caused Subject to be discontinued from the study? |
|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>DDMMMYYYY/HH:MM (X) | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXX | xx | XX | XX/<br>XXX | xx |
| XXXXX | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>Ongoing | XXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXX | Yes: XXXXXX | XXX | XX/<br>XXX | XXX |
| | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/HH:MM (X) /<br>DDMMMYYYY/HH:MM (X) | XXXXXXXXX/<br>XXXXXXXX/<br>XXXXXXXX | XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXX | XX | XX | XX/<br>XXX | XX |

Abbreviations: AESI = adverse event of special interest; COVID-19 = coronavirus 2019; DMR = duodenal mucosal resurfacing; GI = gastrointestinal; MedDRA = medical dictionary for regulatory activities; TEAE = treatment emergent adverse event; UADE = unanticipated adverse device effect.

Note: Study day is calculated relative to the date of index procedure. Adverse events were coded using MedDRA version 22.0. A TEAE is any AE that starts or worsens after the start of DMR or Sham procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If time missing, display "- -:- -". If Other Action Taken? is Other or Concomitant Medication, concatenate all specify fields with a semicolon. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." Ensure correct MedDRA version is printed in footnote.

<sup>[2]</sup> COVID-19 related AEs include the following MedDRA preferred terms:





#### Listing 16.2.7.1 (cont.) Adverse Events All Subjects

| | Randomized<br>Treatment<br>[1] | System Organ Class<br>Preferred Term/<br>Verbatim Term | Start Date/Time<br>/ (Study Day)/<br>End Date/Time (Study<br>Day) | AESI? | Time from<br>DMR/Sham<br>Procedure<br>(Days,<br>Hours) | Duration<br>of<br>Episode<br>(Days,<br>Hours) | n<br>If Diarrhea,<br>Characteristics/Other<br>Clinical Symptoms | If GI Bleeding,<br>Add'I Lab or<br>Diagnostic<br>Tests<br>Conducted? | Cause for<br>Fever/Add'l<br>Symptoms | Other<br>Additional<br>Symptoms | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXX | XXXXXXXXXXXXX | C/DDMMMYYYY/HH:MM<br>C(X)/<br>DDMMMYYYY/HH:MM<br>(X) | | XX, XX | XX, XX | XXXXX/XXXXX | xx | xxxxx/xxxxx | xxxxx | XX |
| XXXXX | XXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | )Ongoing | XXX;XXXXX | XXX, XX | XX, XX | xxxxx | XXX | XXXXX | xxxxx | XX |
| | XXXXX | | (/DDMMMYYYY/HH:MM<br>((X)<br>DDMMMYYYY/HH:MM | | XX, XX | XX, XX | XXXXX/XXXX | XX | XXXXX/XXXX | XXXXX | XX |

Abbreviation: AESI = adverse event of special interest; COVID-19 = coronavirus 2019; DMR = duodenal mucosal resurfacing; GI = gastrointestinal; TEAE = treatment emergent adverse event; UADE = unanticipated adverse device effect.

Note: Study day is calculated relative to the date of index procedure. Adverse events were coded using MedDRA version 22.0. A TEAE is any AE that starts or worsens after the start of DMR or Sham procedure.

[2] COVID-19 related AEs include the following MedDRA preferred terms:

**Programming note:** Ensure proper MedDRA version is displayed in footnote. If diarrhea other clinical symptoms or if fever addition symptoms is Other, concatenate specify field with a semicolon. Include the PTs upon AE review prior to lock.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.7.2 Hypoglycemia Form All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | FPG >220<br>mg/dL through<br>Week 12 or<br>FPG > 200<br>mg/dL Week<br>12-24? | Reporting<br>Type /<br>Fasting? | FPG #1 Value<br>(unit) / Date (Study<br>Day) | FPG #2 Value<br>(unit) / Date<br>(Study Day) | Clinic Lab<br>Value (unit) /<br>Date (Study<br>Day) | Fasting for Clinic<br>Lab Value? | Rescue<br>Criteria<br>Met? | Rescue<br>Medication<br>Started? | Was<br>Rescue<br>Medication<br>a GLP-1? | Nausea? / Vomiting? / Pre- Existing Diarrhea? | Additional<br>Symptoms? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | xxxxx | XXX | XXXXXXX<br>/ XX | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XX | XX / XX /<br>XX | xxxxx |
| XXXXXX | XXXXXX | XX;XXXXXXX | XXXXXXX<br>/ XXX | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXXXX (xxx)<br>DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XX | XX / XX /<br>XX | XXXXXX |

Abbreviations: DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose; SAE = serious adverse event.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If rescue medication was not started, concatenate the Why field with a semicolon. If rescue medication was not a GLP-1, concatenate reason with a semicolon. Concatenate the specify and other additional symptom fields with a semicolon in the cell.





#### Listing 16.2.8.1.1 Laboratory Data: Complete Blood Count All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | Parameter (unit) | Study<br>Visit | Date of<br>Collection<br>(Study Day) | Standard<br>Results | Change<br>from<br>Baseline<br>[3] | Reference<br>Range<br>[4] | Reference<br>Range Flag | Accession<br>Number | Abnormally<br>Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXX | Hematocrit (unit) | xxxxxx | DDMMMYYYY<br>(X) | XX | | XX – YY | | xxxxxx | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | XXX | XXXXXXX | XX |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXXX | |
| | | | XXXXXX | (X) | ND | | | | | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX | XX – YY | | XXXXXXX | |

Abbreviations: A = abnormal; DMR = duodenal mucosal resurfacing; H = high; L = low. Note: Study day is calculated relative to the date of index procedure.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

<sup>[2]</sup> Baseline is the last measurement taken before the index procedure.

<sup>[3]</sup> Reference range is used to identify potentially clinically significant laboratory values.





Listing 16.2.8.1.2 Laboratory Data: Blood Chemistry All Subjects

Same shell as 16.2.8.1.1

Listing 16.2.8.1.3 Laboratory Data: Urinalysis All Subjects

Same shell as 16.2.8.1.1





#### Listing 16.2.8.1.4 Urine Pregnancy Test All Subjects

| Subject ID | Randomized<br>Treatment [1] | Was Sample Collected? | Collection Date<br>(Study Day) | Result |
|---|---|---|---|---|
| XXXXXX | xxxxxx | XXX | DDMMMYYYY (XX) | XXXXXXX |
| xxxxxx | XXXXXX | xx;xxxxxxx | DDMMMYYYY (XX) | XXXXXXX |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If a sample was not collected, concatenate reason in the cell with a semicolon.





# Listing 16.2.8.1.5 Self Monitoring Blood Glucose and Glycemia Diary All Subjects

| Subject ID | Randomized<br>Treatment [1] | Study Visit | Assessment Date/Time<br>(Study Day) | Timepoint | Was Assessment<br>Performed? | Blood<br>Glucose<br>Result<br>(mg/dL) | Were<br>OADs<br>Taken? | Was<br>Subject<br>Fasting? |
|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | XXXXXXX | DDMMMYYYY / HH:MM<br>(XX) | XXXXXXX | XXX | XXXXXXX | XXX | XXX |
| XXXXXX | xxxxx | XXXXXXX | DDMMMYYYY / HH:MM<br>(XX) | xxxxxx | XX; XXXXXX | XXXXXXX | XXX | XXX |

Abbreviation: DMR = duodenal mucosal resurfacing; OAD = oral antidiabetic medication.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If an assessment was not performed or if OADs were not taken, concatenate reason in the cell with a semicolon. Data from the BDG4 case report form will be the Pre-Breakfast and Pre-Dinner Assessments.





Listing 16.2.8.2 Vital Signs All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | Parameter (unit) | Study<br>Visit | Date of<br>Measurements<br>(Study Day) | Standard<br>Results | Change from<br>Baseline [2] |
|---|---|---|---|---|---|---|
| XXXXX | XXXXX | Weight (kg) | XXXXXX | DDMMMYYYY | XX | |
| | | | | (X) | | |
| | | | XXXXXX | DDMMMYYYY<br>(X) | XX | XX |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

Programming note: Parameters include: Height (cm), Weight (kg), BMI (kg/m²), Pulse Rate (bpm), Sitting Systolic BP (mmHg), Sitting Diastolic BP .mmHg)

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

<sup>[2]</sup> Baseline is the last measurement taken before the index procedure.





#### Listing 16.2.8.3 12-Lead Electrocardiogram (ECG) Results All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was ECG<br>Performed? | Date/Time of<br>ECG<br>(Study Day) | RR<br>Interval<br>(bpm) | Ventricular<br>Rate<br>(bpm) | PR<br>Interval<br>(bpm) | QRS<br>Interval<br>(msec) | QTc<br>Interval<br>(msec) | QTcB<br>Interval<br>(msec) | Overall<br>Interpretation | Abnormality | Significance of Finding |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | xxx | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXX | | |
| | | XX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXXXXX | XXXXXX | XXXXX |
| | | XXX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXXX | | |
| | | XXX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXX | | |
| | | XXX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | xxxxxxxxxx | | |
| | | XX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXXX | | |
| | | XXX | ND ` ´ | | | | | | | | | |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY/<br>HH:MM (XX) | XXX | XXX | XXX | XXX | XXX | XXX | XXXXXXX | | |
| | | XXX | DDMMMYYYY/<br>HH:MM (XX) | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXXXXXXXX | | |

Abbreviations: CS = clinically significant; DMR = duodenal mucosal resurfacing; NCS = not clinically significant; ND = not done. Note: Study day is calculated relative to the date of index procedure.

Programming note: If ECG was not performed, concatenate with reason.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.8.4 MRI Enterography (MRE) All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was MRE<br>Done? | Study<br>Visit | Date/Time of MRE<br>(Study Day) | Clinically Relevant Abnormal Findings? | Test Name | Result |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | XXXXXX | DDMMMYYYY / HH:MM (XX) | XXXXXXX | Scan Evaluable Duodenum Distended Duodenal Wall Thickness Measurement Duodenal Wall Thickening Duodenal Wall Enhancement Duodenal Wall Enhancement Description Duodenal Wall Edema Mucosal Hypoenhancement Delayed Hyperenhancement Duodenal Wall Restricted Diffusion Luminal Narrowing Active Inflammation of Fibrosis Periduodenal Edema and Inflammatory Changes Severe Periduodnal Inflammatory Changes | Y/N Y/N Y/N XX.X Y/N Y/N XXXXXX Y/N Y/N Y/N Y/N |
| | | | | | | Periduodenal Fluid Collections<br>Safety Monitoring Findings | Y/N<br>Y/N |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





Listing 16.2.8.5.1 Lifestyle Counseling All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was Lifestyle Counseling Performed? | Study<br>Visit | Date of<br>Performed<br>(Study Day) | Compliant with Diabetic Diet? | Compliant with Lifestyle and Exercise? | Compliant with Diabetics Medications? |
|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | xxx | xxxxx | DDMMMYYYY<br>(XX) | xxxxxx | xxxxxx | xxxxxxx |

Abbreviation: DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





#### Listing 16.2.8.5.2 Lifestyle Evaluation All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Study<br>Visit | AEs Since<br>Last Visit? | Glycemia Diary<br>Reviewed? | Glycemic Events<br>Since Last Visit? | Change in<br>Medications Since<br>Last Visit? | Change in Non-Study<br>Surgical Treatment Since<br>Last Visit? | Instructed to Continue OAD Medication w/o Changes in Regimen? |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | xxxxxx | XX | XX | XXXXXXX | XX | XX | XXX; XXXXX |

Abbreviations: AE = adverse event; DMR = duodenal mucosal resurfacing.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If subject was not instructed to continue anti-diabetic medication without any changes in the prescribed regimen until the Visit 3 procedure, concatenate the reason not instructed with a semicolon.





### Listing 16.2.8.6 Prior and Concomitant Medications All Subjects

| Subject<br>ID | Randomized<br>Treatment [1] | Prior/<br>Concomitant<br>[2] | ATC Class (Level 4)/<br>Preferred Term (ATC Level 5)/<br>Verbatim Term | Type of Medication<br>or Therapy/<br>Indication | Start Date (Study Day)/<br>Stop Date (Study Day) | Dose (unit) | Route | Frequency |
|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXX | Prior | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX | MMMYYYY (-XX)/<br>DDMMMYYYY (-X) | XXXX unit | XXXXXXXX | XXXXX |
| | | Both | XXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXXXXX | XXXXX | MMMYYYY (-X)/<br>Ongoing | XXXX unit | XXXXXXXX | XXXXX |
| | | Concomitant | XXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxx | DDMMMYYYY (X)/<br>DDMMMYYYY (XX) | XXXX unit | XXXXXXXX | XXXXX |

Abbreviations: ATC = anatomic therapeutic chemical; DMR = duodenal mucosal resurfacing; N/A = Not applicable; WHO-DD = World Health Organization drug dictionary. Note: Study day is calculated relative to the date of index procedure. Medications were coded using WHO-DD version March 2019.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment. [2] Prior medications are all medications (including diabetic medications, rescue medications, and non-drug therapies) that were started before the index procedure. Concomitant medications are all medications (including diabetic medications, rescue medications, and non-drug therapies) that were continuing or starting after the index procedure. Both indicates medication that was started prior to the index procedure and continued after the index procedure.

**Programming note:** Concatenate specify field for indication. If Dose unit, Route or Frequency is Other, display other specify text only (i.e., do not display "Other: XXXXXX" but just "XXXXXX"). Sort by subject, start date/time, end date/time, ATC level 4 & PT. Ensure proper WHO-DDE version is printed in footnote.





#### Listing 16.2.8.7.1 Physical Examination All Subjects

| Subject ID | Randomized<br>Treatment [1] | Was Physical Exam<br>Performed? | Exam Date<br>(Study Day) | Body System | Result | If Abnormal,<br>Describe | Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | XXX | DDMMMYYYY (XX) | XXXXXXX | Normal | | |
| 700000 | 700000 | XX | DDMMMYYYY (XX) | XXXXXXXXXXX | Abnormal | XXXXXXXXXXX | XX |
| | | XXX | DDMMMYYYY (XX) | XXXXXXXX | XXXXXXXX | | |
| | | XXX | DDMMMYYYY (XX) | XXXXXXX | XXXXXXXX | | |
| | | XXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXXX | | |
| | | XX | DDMMMYYYY (XX) | XXXXXXXX | XXXXXXXX | | |
| | | XXX | ND ` ´ | | Not Done | | |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY (XX) | XXXXXXXXXXX | XXXXXXXX | | |
| | | XXX | DDMMMYYYY (XX) | XXXXXXXXXX | XXXXXXXX | | |

Abbreviations: DMR = duodenal mucosal resurfacing; ND = not done.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





Listing 16.2.8.7.2
Targeted Physical Examination
All Subjects

#### Same shell as 16.2.8.7.1.

**Programming note:** Body Systems will be: Fundoscopic exam, thyroid palpation, abdominal exam, heart and lung, deep tendon reflex and sensation skin. Add a column before 'Was Physical Exam Performed' labeled 'Reported Signs or Symptoms Since Last Visit.'





Listing 16.2.8.8.1 Patient Contact All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Did Subject<br>Contact<br>Site? | Date of<br>Contact<br>(Study Day) | Experienced 2 or More Occurrences of Hypoglycemia? | Was Diary<br>Reviewed? | Was a Follow-<br>Up Visit<br>Scheduled? /<br>Date of Visit<br>(Study Day) | Clinic Lab<br>Value (FPG)<br>(unit) / Clinical<br>Lab Value<br>Date<br>(Study Day) | Was<br>Subject<br>Fasting? | Were<br>Changes<br>in<br>Medication<br>Made? | Any<br>other<br>Action<br>Taken? | Experienced an AE/SAE? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXX | DDMMMYYYY<br>(XX) | XXX | xxx | XXX /<br>DDMMMYYYY<br>(XX) | XXXXXXX<br>(xxx) /<br>DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XXX | DDMMMYYYY<br>(XX) | XXX | XX; | XXX /<br>DDMMMYYYY<br>(XX) | XXXXXXX<br>(xxx) /<br>DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XXX |

Abbreviation: AE = adverse event; DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose; SAE = serious adverse event. Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** If no changes in medication were made, concatenate reason in the cell with a semicolon.





#### Listing 16.2.8.8.2 Day 7 Telephone Contact All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was the<br>Subject<br>Contacted<br>by<br>Phone? | Date of<br>Contact<br>(Study Day) | Experience<br>Hypoglycemic<br>Events Since<br>Discharge? | Experience<br>FPG meeting<br>Hypoglycemic<br>Rescue<br>Threshold<br>Since<br>Discharge? | Experience<br>AEs Since<br>Discharge? | Pre-<br>Planned<br>Non-Study<br>Surgical<br>Treatment<br>Since Last<br>Call? | Change in<br>Medication<br>Since<br>Discharge? | Compliant<br>with Post-<br>Procedure<br>Diet Over<br>Last 7<br>Days? | Reminded<br>About<br>Specific<br>14 Day<br>Post-<br>Procedure<br>Diet? | Provided Instructions and Reminded to conduct Blood Glucose Monitoring 4x per Day for 7 Days? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XXX;<br>XXXXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | XXXXXXX | DDMMMYYYY<br>(XX) | XXX | XXX | XX | XX | XXX | xxx | XXX | XXX |

Abbreviation: AE = adverse event; DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** if the subject was not contacted by phone, concatenate reason with a semicolon. If the subject had pre-planned non-study surgical treatment, concatenate specify field in the cell with a semicolon.





# Listing 16.2.8.8.3 Day 14 Telephone Contact All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was the<br>Subject<br>Contacted<br>by Phone? | Date of<br>Contact<br>(Study Day) | Experience<br>Hypoglycemic<br>Events Since<br>Day 7 Call? | Experience<br>FPG<br>Meeting<br>Rescue<br>Threshold<br>Since Day<br>7 Call? | Experience<br>AEs Since<br>Day 7<br>Call? | Pre-Planned<br>Non-Study<br>Surgical<br>Treatment<br>Since Day 7<br>Call? | Change in<br>Medication<br>Since Day 7<br>Call? | Compliant<br>with Post-<br>Procedure<br>Diet Over<br>Last 7<br>Days? | Reminded<br>to Start<br>Standard<br>Diabetic<br>Diet and<br>Exercise? | Reminded<br>to Measure<br>Blood<br>Sugar and<br>Complete<br>the<br>Glycemia<br>Diary? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XXX;<br>XXXXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX | XX | XX | XXX | XXX | XXX | XXX |

Abbreviation: AE = adverse event; DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** if the subject was not contacted by phone, concatenate reason with a semicolon. If the subject had pre-planned non-study surgical treatment, concatenate specify field in the cell with a semicolon.





Listing 16.2.8.8.4 Telephone Contact All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was the<br>Subject<br>Contacted<br>by Phone? | Date of<br>Contact<br>(Study Day) | Experience<br>Hypoglycemic<br>Events Since<br>Last Visit? | Experience<br>FPG<br>Meeting<br>Rescue<br>Threshold<br>Since<br>Discharge | Experience<br>AEs Since<br>Last Visit? | Pre-Planned<br>Non-Study<br>Surgical<br>Treatment<br>Since Last<br>Call? | Change in<br>Medication<br>Since Last<br>Visit? | Compliant<br>with<br>Standard<br>Diet Since<br>Last<br>Visit? | Was<br>Lifestyle<br>Counseling<br>Provided? | Reminded<br>to Measure<br>Blood<br>Sugar and<br>Complete<br>the<br>Glycemia<br>Diary? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX | XXX | XXX;<br>XXXXXX | XXX | XXX | XXX | XXX |
| XXXXXX | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX | XX | XX | XXX | XXX | XXX | xxx |

Abbreviation: AE = adverse event; DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose.

Note: Study day is calculated relative to the date of index procedure.

[1] Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.

**Programming note:** if the subject was not contacted by phone, concatenate reason with a semicolon. If the subject had pre-planned non-study surgical treatment, concatenate specify field in the cell with a semicolon.





#### Listing 16.2.8.8.5 Follow Up Office Visit All Subjects

| Subject<br>ID | Randomized<br>Treatment<br>[1] | Was the<br>Follow Up<br>Office Visit<br>Performed? | Date of Visit<br>(Study Day) | Experience Hypoglycemic Events / FPG Meeting Rescue Threshold / AEs Since Last Call? | Pre-<br>Planned<br>Non-<br>Study<br>Surgical<br>Treatment<br>Since<br>Last Call? | Change in<br>Medication<br>Since Last<br>Call? | Compliant with Prescribed Diabetes Medications / Diabetic Diet / Lifestyle and Exercise Since Last Call? | Was<br>Lifestyle<br>Counseling<br>Provided? | Reminded to Measure Blood Sugar and Complete Diary / Maintain Diabetes Medication Regimen? | Which<br>Treatment<br>Does<br>Subject<br>Think<br>He/She<br>Received? | How<br>Confident<br>is the<br>Subject<br>of the<br>Guess? | What<br>are the<br>Reasons<br>for This<br>Guess? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | XXXXXX | xxxxxx | DDMMMYYYY<br>(XX) | XXX | XXX;<br>XXXXXX | XXX | XXX / XXX /<br>XXX | xxx | XXX | XXX | XXX | xxx |
| XXXXXX | xxxxxx | XXXXXXX | DDMMMYYYY<br>(XX) | xxx | XX | XXX | XXX / XXX /<br>XXX | XXX | XXX | XXX | XXX | xxx |

Abbreviation: AE = adverse event; DMR = duodenal mucosal resurfacing; FPG = fasting plasma glucose.

Note: Study day is calculated relative to the date of index procedure.

**Programming note:** if the follow up office visit was not performed, concatenate reason with a semicolon. If the subject had pre-planned non-study surgical treatment, concatenate specify field in the cell with a semicolon.

<sup>[1]</sup> Subjects were randomized to either DMR or Sham procedure in the double-blind period. After Week 24, Sham subjects had the opportunity to crossover and receive DMR treatment.





### 14.4. Planned Figure Shells

Not Applicable.



### **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|---------------------------------|
| AE | Adverse event |
| AESI | Adverse events special interest |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| AT | As treated |
| ATC | Anatomical therapeutic chemical |
| BMI | Body mass index |
| CEC | Central ethics committee |
| CFR | Code of federal regulations |
| CI | Confidence intervals |
| COVID-19 | Coronavirus 2019 |
| CRF | Case report form |
| CS | Clinically significant |
| CSR | Clinical study report |
| DBP | Diastolic blood pressure |
| DMC | Data monitoring committee |
| DMR | Duodenal Mucosal Resurfacing |
| EC | Ethics committee |
| ECG | Electrocardiogram |



| Abbreviation | Definition |
|--------------|----------------------------------------------|
| eCRF | Electronic case report form |
| EMA | European medicines agency |
| EU | European Union |
| FDA | Food and drug administration |
| FPG | Fasting plasma glucose |
| GCP | Good clinical practice |
| HbA1c | Hemoglobin A1c |
| HR | Heart rate |
| IC or ICF | Informed consent or informed consent form |
| ICH | International council for harmonization |
| ID | Identification |
| IQR | Interquartile range |
| ITT | Intent-to-treat |
| MedDRA | Medical dictionary for regulatory activities |
| MMRM | Mixed effect model repeat measurement |
| MRE | Magnetic resonance imaging enterography |
| N | Number |
| NA | Not applicable |
| NCS | Non-clinically significant |
| OAD | Oral antidiabetic medication |
| PD | Protocol deviation |



| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| PE | Physical examination |
| PI | Principal investigator |
| PROMIS | Patient-Reported Outcomes Measurement Information |
| QOL | Quality of life |
| RR | Respiratory rate or relative rate |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS® | A software system used for data analysis |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SF | Screen failure |
| SF-36 | Short Form Health Survey (36) |
| SOC | System organ class |
| T2D | Type II Diabetes |
| TEAE | Treatment-emergent adverse event |
| UACR | Urine Albumin-to-Creatinine Ratio |
| UADE | Unanticipated adverse device effect |
| US | United States |
| USA | United States of America |
| WHO | World health organization |
| WHO-DD | World health organization drug dictionary |



